CLINICAL TRIAL: NCT03746015
Title: An Open-Label, Phase 2 Trial to Investigate the Humoral and Cell-Mediated Immune Responses and Safety of a Tetravalent Dengue Vaccine Candidate (TDV) Administered Subcutaneously in Flavivirus-Naïve and Dengue-Immune Healthy Adults
Brief Title: Immunogenicity and Safety of Tetravalent Dengue Vaccine Candidate (TDV) in Flavivirus-Naïve and Dengue-Immune Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEN-210
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Dengue Fever
Keywords: Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TDV: Flavivirus-naïve (Experimental): Tetravalent Dengue Vaccine (TDV) 0.5 mL, subcutaneous (SC) injection, once on Day 1 (first dose) and then on Day 90 (second dose). Participants who were flavivirus-naïve were included in this group.
  Interventions: Biological: TDV
- TDV: DENV Immune: DENV-1 Positive (Experimental): TDV 0.5 mL, SC injection, once on Day 1 (first dose) and then on Day 90 (second dose).
  Participants with serology consistent with primary infection by wild type dengue virus serotype-1 (DENV-1) were included in this group.
  Interventions: Biological: TDV
- TDV: DENV Immune: DENV-3 Positive (Experimental): TDV 0.5 mL, SC injection, once on Day 1 (first dose) and then on Day 90 (second dose).
  Participants with serology consistent with primary infection by DENV-3 were included in this group.
  Interventions: Biological: TDV

INTERVENTIONS:
Biological: TDV — TDV subcutaneous injection comprised of 1 molecularly characterized, attenuated dengue virus strain, and 3 chimeric dengue virus strains with potencies of not less than 3.3, 2.7, 4.0, and 4.5 log10 plaque forming units (PFU) per dose of TDV-1, TDV-2, TDV-3, and TDV-4, respectively.

SUMMARY:
The purpose of this study is to assess the neutralizing antibody response against each dengue serotype post-vaccination.

DETAILED DESCRIPTION:
The vaccine being tested in this study is Takeda's Tetravalent Dengue Vaccine Candidate (TDV). TDV is being tested to protect people against dengue fever. This study will look at the immunogenicity and safety of TDV in flavivirus-naïve and dengue-immune adults.

The study will enroll approximately 44 patients. Participants will be categorized into two groups based on results from serological testing performed by the trial center outside the scope of this trial (up to 70 days [10 weeks] prior to Day 1 [Month 0]):

Group 1: Flavivirus-Naïve Participants Group 2: Dengue-Immune Participants

All participants will receive subcutaneous injection of TDV on Day 1 (Month 0) and Day 90 (Month 3).

This trial will be conducted in the United States. The overall time to participate in this study is 12 months. Participants will make multiple visits to the clinic, and 9 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
2. Group 1 only: immunologically naïve to dengue, Zika, Yellow Fever (YF), Japanese Encephalitis (JE), West Nile (WN) (based on negative results for detection of anti-DENV, anti-Zika, anti-YF, anti-JE, anti-WN antibodies) as documented by serological testing performed by the trial center outside the scope of this trial (up to 70 days [10 weeks] prior to Day 1 [Month 0]).
3. Group 2 only: serology consistent with primary infection with either DENV-1 or DENV-3 (defined as detectable neutralizing antibodies against DENV-1 or DENV-3 only, or titers for DENV-1 or DENV-3 ≥4-times higher than titers for the 2 other dengue serotypes) as documented by serological testing performed by the trial center outside the scope of this trial (up to 70 days [10 weeks] prior to Day 1 [Month 0]).

Exclusion Criteria:

1. Has clinically active significant infection (as assessed by the investigator) or body temperature ≥38°C (100.4°F) within 3 days of the intended date of vaccination.
2. Has history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (eg, Guillain-Barré syndrome).
3. Known or suspected impairment/alteration of immune function including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks and/or ≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks and/or ≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0).
   3. Administration of immunoglobulins and/or any blood products within 3 months prior to Day 1 (Month 0) or planned administration during the trial.
   4. Receipt of immunostimulants within 60 days prior to Day 1 (Month 0).
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (Month 0).
   6. Known Human Immunodeficiency Virus (HIV) infection or HIV-related disease.
   7. Hepatitis C virus infection.
   8. Genetic immunodeficiency.
4. Has planned vaccination (during the trial conduct) against any non-dengue flavivirus (eg, Zika, YF, JE, WN, tick-borne encephalitis, or Murray-Valley encephalitis).
5. Planned travel (during the trial conduct) to any area endemic for dengue.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Optimal Research, Peoria, Illinois
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 28 December 2018 to 1 March 2021.
Pre-assignment Details: Healthy participants were enrolled in this study to receive Tetravalent Dengue Vaccine (TDV) on Days 1 and 90. One participant did not meet the randomization criteria and was not allocated to any of the pre-defined study groups and was excluded from all analyses except safety analysis.
Period: Overall Study
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Started | 22 | 4 | 3
Safety Population (Safety Analysis Set included all participants who received at least one dose of trial vaccine. One participant was seropositive for all dengue strains at Screening and was therefore not allocated to dengue serotype 1 or 3 positive groups. The participant did receive two vaccine doses and was thus included in Safety Analysis Set.) | 22 | 4 | 3
Completed | 21 | 4 | 3
Not Completed | 1 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of trial vaccine and for whom a valid pre-dose and at least one valid post-dose blood sample was taken.
Groups:
- TDV: Flavivirus-naïve: TDV 0.5 mL, SC injection, once on Day 1 (first dose) and then on Day 90 (second dose).
  Participants who were flavivirus-naïve were included in this group.
- TDV: DENV Immune: DENV-1 Positive: TDV 0.5 mL, SC injection, once on Day 1 (first dose) and then on Day 90 (second dose).
  Participants with serology consistent with primary infection by DENV-1 were included in this group.
- Total: Total of all reporting groups
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Total
Number analyzed (Participants) | 21 | 4 | 3 | 28
Age, Continuous [Mean (Full Range); unit: years] | 33.57 [22.0 to 58.0] | 42.25 [32.0 to 53.0] | 35.00 [33.0 to 38.0] | 34.96 [22 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 0 | 12
  Male | 11 | 2 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 3 | 3 | 27
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 17 | 3 | 1 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 4 | 3 | 28
Height [Mean (Full Range); unit: centimeter (cm)] | 169.18 [148.6 to 182.1] | 175.01 [163.6 to 188.0] | 174.33 [172.7 to 176.3] | 170.56 [148.6 to 188]
Weight [Mean (Full Range); unit: kilogram (kg)] | 71.54 [48.7 to 101.2] | 71.86 [64.9 to 78.0] | 79.15 [68.0 to 97.8] | 72.4 [48.7 to 101.2]
Body Mass Index (BMI) [Mean (Full Range); unit: kilogram per meter square (kg/m^2)] — BMI= weight (kg)/height (m^2)
  kilogram per meter square (kg/m^2) | 24.74 [19.4 to 32.0] | 23.48 [20.4 to 25.2] | 25.90 [22.7 to 31.4] | 24.68 [19.4 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 15
Description: GMT of neutralizing antibodies were measured for each of the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by microneutralization test 50% (MNT50).
Time Frame: Day 15
Population: Per Protocol Set (PPS) included all participants in the Full Analysis Set (FAS) who had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
titer
  DENV-1 | 58.9 [28.9 to 120.0] | 15325.2 [32.4 to 7241076.9] | 5510.0 [1271.4 to 23879.4]
  DENV-2 | 11.2 [6.5 to 19.2] | 5200.2 [13.9 to 1947484.8] | 4142.7 [694.3 to 24718.0]
  DENV-3 | 42.1 [16.2 to 109.8] | 2468.7 [0.0 to 272077002.4] | 7244.0 [5083.2 to 10323.3]
  DENV-4 | 19.7 [10.6 to 36.7] | 1996.4 [0.5 to 8424572.5] | 4909.2 [2503.2 to 9628.0]

2. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 30 (Month 1)
Description: GMT of neutralizing antibodies were measured for each of the four dengue serotypes: DENV-1, DENV-2, DENV-3, and DENV-4, by MNT50.
Time Frame: Day 30 (Month 1)
Population: PPS included all participants in the FAS who had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
titer
  DENV-1 | 336.1 [168.8 to 669.3] | 45437.3 [58.0 to 35607948.4] | 11091.9 [706.7 to 174081.3]
  DENV-2 | 11557.1 [6408.8 to 20841.2] | 12317.0 [2677.3 to 56665.6] | 12221.9 [1004.9 to 148651.5]
  DENV-3 | 344.7 [146.3 to 812.6] | 7273.6 [2983.8 to 17730.9] | 19062.2 [3584.4 to 101373.6]
  DENV-4 | 141.1 [69.1 to 288.0] | 5094.3 [888.2 to 29218.2] | 5231.1 [2064.2 to 13256.7]

3. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 60 (Month 2)
Description: as for outcome 2
Time Frame: Day 60 (Month 2)
Population: PPS included all participants in the FAS who had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
titer
  DENV-1 | 258.5 [102.0 to 655.4] | 28109.0 [65.7 to 12030804.9] | 7827.8 [1701.7 to 36007.3]
  DENV-2 | 6293.0 [3655.7 to 10833.1] | 9641.1 [4219.1 to 22030.9] | 7236.5 [432.9 to 120961.1]
  DENV-3 | 174.6 [79.7 to 382.9] | 6174.2 [200.8 to 189874.6] | 15536.5 [3282.7 to 73532.6]
  DENV-4 | 78.2 [35.0 to 174.7] | 6122.7 [1974.7 to 18984.1] | 4254.8 [720.8 to 25116.0]

4. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 90 (Month 3)
Description: as for outcome 2
Time Frame: Day 90 (Month 3)
Population: PPS included all participants in the FAS who had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
titer
  DENV-1 | 197.5 [82.7 to 471.7] | 24989.5 [244.4 to 2554755.6] | 8111.3 [2866.7 to 22950.5]
  DENV-2 | 4077.0 [2535.6 to 6555.5] | 9167.4 [4646.6 to 18086.6] | 5450.5 [857.1 to 34661.2]
  DENV-3 | 145.7 [82.0 to 258.9] | 7043.3 [1348.3 to 36792.6] | 10172.1 [3690.3 to 28038.7]
  DENV-4 | 79.2 [37.3 to 168.0] | 3240.2 [9.6 to 1095309.8] | 4372.2 [857.1 to 22304.5]

5. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 105
Description: as for outcome 2
Time Frame: Day 105
Population: PPS included all participants in the FAS who had no major protocol violations. Overall number analyzed are the number of participants with data available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 6 | 1 | 3
titer
  DENV-1 | 326.0 [117.8 to 902.2] | 13354.0 [NA to NA] — The 95% confidence interval (CI) was not estimable due to insufficient number of observations. | 6720.6 [3035.5 to 14879.7]
  DENV-2 | 3784.9 [1419.9 to 10088.5] | 5810.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 5635.6 [1094.4 to 29020.9]
  DENV-3 | 221.0 [55.9 to 873.8] | 2360.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 12835.4 [3232.2 to 50971.0]
  DENV-4 | 211.6 [73.5 to 609.2] | 2181.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 4011.8 [1075.2 to 14969.0]

6. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 120 (Month 4)
Description: as for outcome 2
Time Frame: Day 120 (Month 4)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 12 | 2 | 3
titer
  DENV-1 | 433.8 [149.0 to 1262.8] | 27123.8 [5.1 to 144760235.6] | 9242.2 [3693.4 to 23127.1]
  DENV-2 | 3636.1 [1912.1 to 6914.5] | 7424.1 [1187.8 to 46402.4] | 6187.5 [1220.4 to 31371.1]
  DENV-3 | 132.1 [58.7 to 297.5] | 4179.0 [16.5 to 1060298.0] | 10402.8 [3725.1 to 29051.2]
  DENV-4 | 112.3 [67.4 to 187.3] | 2428.6 [16.2 to 364777.8] | 3835.1 [619.1 to 23755.8]

7. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 150 (Month 5)
Description: as for outcome 2
Time Frame: Day 150 (Month 5)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 15 | 1 | 3
titer
  DENV-1 | 266.7 [125.5 to 566.7] | 15703.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 7652.0 [3152.7 to 18572.6]
  DENV-2 | 2415.2 [1355.6 to 4303.0] | 7081.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 4589.6 [586.8 to 35898.7]
  DENV-3 | 137.0 [76.4 to 245.5] | 2829.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 8627.9 [2944.9 to 25277.7]
  DENV-4 | 120.5 [64.1 to 226.8] | 1729.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 3593.4 [585.2 to 22065.1]

8. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 180 (Month 6)
Description: as for outcome 2
Time Frame: Day 180 (Month 6)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 15 | 2 | 3
titer
  DENV-1 | 194.4 [92.8 to 407.4] | 22880.8 [2540.1 to 206105.7] | 4101.6 [466.2 to 36082.4]
  DENV-2 | 1920.1 [1070.8 to 3443.2] | 10697.4 [138.0 to 829066.2] | 5458.3 [622.8 to 47838.6]
  DENV-3 | 98.2 [55.2 to 174.6] | 4198.3 [601.5 to 29302.7] | 7495.0 [3027.3 to 18556.1]
  DENV-4 | 76.1 [37.9 to 152.8] | 2797.3 [122.6 to 63824.0] | 2742.4 [769.7 to 9770.8]

9. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 270 (Month 9)
Description: as for outcome 2
Time Frame: Day 270 (Month 9)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 11 | 1 | 3
titer
  DENV-1 | 121.7 [23.4 to 631.8] | 16158.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 3913.9 [982.7 to 15587.9]
  DENV-2 | 1584.0 [1038.1 to 2417.1] | 8585.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 3925.6 [520.5 to 29606.8]
  DENV-3 | 85.6 [44.3 to 165.2] | 3727.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 5985.8 [5342.8 to 6706.1]
  DENV-4 | 39.5 [16.8 to 92.9] | 1684.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 2021.3 [400.1 to 10210.5]

10. Primary Outcome: GMT of Neutralizing Antibodies for Each of the Four Dengue Serotypes at Day 360 (Month 12)
Description: as for outcome 2
Time Frame: Day 360 (Month 12)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 11 | 1 | 2
titer
  DENV-1 | 154.6 [36.5 to 655.2] | 17546.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 2623.5 [149.6 to 46022.7]
  DENV-2 | 1287.8 [581.0 to 2854.6] | 9623.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 1523.7 [4.8 to 479413.6]
  DENV-3 | 77.0 [48.2 to 122.9] | 4112.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 5287.8 [613.1 to 45608.8]
  DENV-4 | 29.8 [11.7 to 75.9] | 1171.0 [NA to NA] — The 95% CI was not estimable due to insufficient number of observations. | 1695.3 [92.1 to 31197.8]

11. Secondary Outcome: Percentage of Participants With Interferon-gamma (IFN-γ) Enzyme-linked Immunospot (ELISpot) Responses to Tetravalent Dengue Vaccine (TDV)
Description: IFN-γ ELISpot response >3 times higher compared with baseline (no peptide) and ≥5 spots per 10^6 peripheral blood mononuclear cells (PBMCs) was defined as cellular immune response. Cellular immune response to any peptide pool was reported. The peptide pools included pre-membrane envelope (prME), capsid (C), non-structural proteins (NS): NS1, NS2, NS3, NS4 and NS5 for DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: Days 30 (Month 1), 90 (Month 3), 120 (Month 4), 180 (Month 6), 360 (Month 12)
Population: PPS included all participants in the FAS who had no major protocol violations. Number analyzed is the number of participants with data available for analysis for the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
percentage of participants
  DENV-1 Day 30 (Month 1) | 100 [83.9 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-1 Day 90 (Month 3) | 95.2 [83.2 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-1 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-1 Day 120 (Month 4) | 100 [73.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-1 Day 180 (Month 6): number analyzed (Participants) | 15 | 2 | 3
  DENV-1 Day 180 (Month 6) | 93.3 [68.1 to 99.8] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-1 Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  DENV-1 Day 360 (Month 12) | 90.9 [69.2 to 100] | 100 [2.5 to 100] | 100 [15.8 to 100]
  DENV-2 Day 30 (Month 1) | 100 [83.9 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-2 Day 90 (Month 3) | 100 [83.9 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-2 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-2 Day 120 (Month 4) | 100 [73.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-2 Day 180 (Month 6): number analyzed (Participants) | 15 | 2 | 3
  DENV-2 Day 180 (Month 6) | 100 [78.2 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-2 Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  DENV-2 Day 360 (Month 12) | 100 [71.5 to 100] | 100 [2.5 to 100] | 100 [15.8 to 100]
  DENV-3 Day 30 (Month 1) | 90.5 [69.6 to 98.8] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-3 Day 90 (Month 3) | 85.7 [63.7 to 97.0] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-3 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-3 Day 120 (Month 4) | 100 [73.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-3 Day 180 (Month 6): number analyzed (Participants) | 15 | 2 | 3
  DENV-3 Day 180 (Month 6) | 73.3 [44.9 to 92.2] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-3 Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  DENV-3 Day 360 (Month 12) | 90.9 [58.7 to 99.8] | 100 [2.5 to 100] | 100 [15.8 to 100]
  DENV-4 Day 30 (Month 1) | 76.2 [52.8 to 91.8] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-4 Day 90 (Month 3) | 81.0 [62.1 to 96.8] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-4 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-4 Day 120 (Month 4) | 100 [73.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  DENV-4 Day 180 (Month 6): number analyzed (Participants) | 15 | 2 | 3
  DENV-4 Day 180 (Month 6) | 93.3 [68.1 to 99.8] | 50.0 [1.3 to 98.7] | 100 [29.2 to 100]
  DENV-4 Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  DENV-4 Day 360 (Month 12) | 54.5 [42.1 to 99.6] | 100 [2.5 to 100] | 100 [15.8 to 100]

12. Secondary Outcome: Magnitude of Cellular Immune Response Assessed by Number of Spot Forming Cells [SFC]/10^6 Peripheral Blood Mononuclear Cells (PBMCs) Measured by IFN-γ ELISpot Responses to TDV
Description: The magnitude of cellular immune response was assessed by the number of SFC/10^6 PBMCs. IFN-γ ELISpot response >3 times higher compared with baseline (no peptide) and ≥5 spots per 10^6 PBMCs was defined as cellular immune response. Cellular immune response to any peptide pool was reported. The peptide pools included prME, C, NS1, NS2, NS3, NS4 and NS5 for DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: Days 30 (Month 1), 90 (Month 3), 120 (Month 4), 180 (Month 6), 360 (Month 12)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: SFC/10^6 PBMCs
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
SFC/10^6 PBMCs
  DENV-1 Day 30 (Month 1) | 232.3016 (407.55450) | 2480.0000 (3486.03643) | 301.6667 (159.39992)
  DENV-1 Day 90 (Month 3): number analyzed (Participants) | 20 | 2 | 3
  DENV-1 Day 90 (Month 3) | 189.5834 (350.89563) | 1772.5000 (2485.48034) | 235.0000 (109.65856)
  DENV-1 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-1 Day 120 (Month 4) | 209.8611 (329.52941) | 1517.5000 (2138.99801) | 116.6667 (76.53975)
  DENV-1 Day 180 (Month 6): number analyzed (Participants) | 14 | 2 | 3
  DENV-1 Day 180 (Month 6) | 162.5000 (237.01829) | 1994.1665 (2806.03517) | 242.7777 (166.35251)
  DENV-1 Day 360 (Month 12): number analyzed (Participants) | 10 | 1 | 2
  DENV-1 Day 360 (Month 12) | 235.1667 (340.48572) | 5.0000 (NA) — Standard deviation (SD) was not estimable for a single participant. | 104.1665 (69.53193)
  DENV-2 Day 30 (Month 1) | 1156.9048 (1676.59869) | 1847.5000 (2365.27218) | 551.6667 (309.89245)
  DENV-2 Day 90 (Month 3) | 912.4603 (979.81060) | 1462.5000 (1750.08928) | 352.2223 (267.42243)
  DENV-2 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-2 Day 120 (Month 4) | 999.3056 (1416.74554) | 1237.5000 (1566.24152) | 161.6667 (150.52685)
  DENV-2 Day 180 (Month 6): number analyzed (Participants) | 15 | 2 | 3
  DENV-2 Day 180 (Month 6) | 965.1111 (1154.31464) | 2070.0000 (2807.21392) | 375.5557 (70.56015)
  DENV-2 Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  DENV-2 Day 360 (Month 12) | 974.0909 (1266.49305) | 180.0000 (NA) — Standard deviation (SD) was not estimable for a single participant. | 149.1665 (93.10263)
  DENV-3 Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  DENV-3 Day 30 (Month 1) | 246.5789 (331.14209) | 2035.0000 (2807.21392) | 295.0000 (115.32563)
  DENV-3 Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  DENV-3 Day 90 (Month 3) | 184.8148 (273.48687) | 215.0000 (282.84271) | 226.1113 (212.99673)
  DENV-3 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-3 Day 120 (Month 4) | 156.1112 (280.56878) | 1565.0000 (2192.03102) | 353.3333 (158.61379)
  DENV-3 Day 180 (Month 6): number analyzed (Participants) | 11 | 2 | 3
  DENV-3 Day 180 (Month 6) | 164.0909 (233.54441) | 1726.6665 (2413.59091) | 120.5553 (132.31197)
  DENV-3 Day 360 (Month 12): number analyzed (Participants) | 10 | 1 | 2
  DENV-3 Day 360 (Month 12) | 137.6666 (194.74138) | 5.0000 (NA) — Standard deviation (SD) was not estimable for a single participant. | 123.3335 (16.49892)
  DENV-4 Day 30 (Month 1): number analyzed (Participants) | 16 | 2 | 3
  DENV-4 Day 30 (Month 1) | 224.0625 (420.90109) | 395.0000 (473.76154) | 153.3333 (219.10804)
  DENV-4 Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  DENV-4 Day 90 (Month 3) | 153.0392 (290.81317) | 362.5000 (477.29708) | 71.6667 (38.11558)
  DENV-4 Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  DENV-4 Day 120 (Month 4) | 172.6388 (373.16791) | 57.5000 (74.24621) | 160.0000 (205.36553)
  DENV-4 Day 180 (Month 6): number analyzed (Participants) | 14 | 1 | 3
  DENV-4 Day 180 (Month 6) | 162.2619 (378.98856) | 573.3330 (NA) — Standard deviation (SD) was not estimable for a single participant. | 155.0000 (165.86485)
  DENV-4 Day 360 (Month 12): number analyzed (Participants) | 6 | 1 | 2
  DENV-4 Day 360 (Month 12) | 215.0000 (325.02308) | 40.0000 (NA) — Standard deviation (SD) was not estimable for a single participant. | 75.8335 (62.46086)

13. Secondary Outcome: Phenotype Characterization of Cellular Immune Response to TDV Assessed as Percentage of Total CD4+ T Cells by Intracellular Cytokine Staining (ICS)
Description: Phenotype characterization of cellular immune response was performed in a subset of participants with IFN- γ ELISPOT responses >50 SFC/10^6 cells and availability of sufficient cells. Markers included cluster of differentiation (CD) 4, CD8, IFN-γ, tumor necrosis factor-alpha (TNF-α) and interleukin-2 (IL-2). The peptide pools included C, NS1, NS2/4, NS3, NS5 for DENV-2 and prME for DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: Days 15, 30 (Month 1), 90 (Month 3), 105, 120 (Month 4), and 360 (Month 12)
Population: Intracellular Cytokine Staining (ICS) Subset included participants from PPS (all participants in the FAS who had no major protocol violations) who had IFN-γ ELISPOT responses > 50 SFC/10^6 PBMCs and availability of sufficient cells for analysis. Number analyzed is the number of participants with data available for analysis for the specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T cells
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
percentage of CD4+ T cells
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 15 | 0.0039595 (0.00434343) | 0.0190000 (0.01272792) | 0.0010800 (0.00175923)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0040266 (0.00433388) | 0.0235670 (0.03188062) | 0.0042860 (0.00392989)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0022368 (0.00317381) | 0.0023500 (0.00332340) | 0.0013000 (0.00162631)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 105 | 0.0013760 (0.00241658) | 0.0024200 (NA) — SD was not estimable for a single participant. | 0.0005800 (0.00100459)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0027200 (0.00460175) | 0.0108200 (0.00950352) | 0.0039300 (0.00413312)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0023000 (0.00188396) | 0.0025300 (NA) — SD was not estimable for a single participant. | 0.0019185 (0.00261842)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 15 | 0.0015836 (0.00205944) | 0.0017250 (0.00023335) | 0.0010800 (0.00175923)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1) | 0.0028357 (0.00490865) | 0.0029000 (0.00410122) | 0.0008220 (0.00084058)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3) | 0.0010256 (0.00147028) | 0.0000000 (0.00000000) | 0.0005700 (0.00098727)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 105 | 0.0010760 (0.00089456) | 0.0000600 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4) | 0.0018854 (0.00346501) | 0.0006950 (0.00098288) | 0.0009263 (0.00157941)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12) | 0.0005916 (0.00126206) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 15 | 0.0024555 (0.00404542) | 0.0196200 (0.02214658) | 0.0061433 (0.00488514)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0023374 (0.00257822) | 0.0230380 (0.03247317) | 0.0075220 (0.00887617)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0006646 (0.00100992) | 0.0077600 (0.01097430) | 0.0049000 (0.00652393)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 105 | 0.0036640 (0.00370999) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0069667 (0.01073570)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0015773 (0.00239811) | 0.0087700 (0.01240265) | 0.0031500 (0.00279426)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0004526 (0.00059075) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0024485 (0.00167089)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 15 | 0.0027775 (0.00490646) | 0.0013760 (0.00084004) | 0.0132000 (0.00930161)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 30 (Month 1) | 0.0034686 (0.00432300) | 0.0065550 (0.00927017) | 0.0021460 (0.00082412)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 90 (Month 3) | 0.0012968 (0.00161555) | 0.0055000 (0.00777817) | 0.0011827 (0.00198127)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 105 | 0.0015260 (0.00124341) | 0.0018300 (NA) — SD was not estimable for a single participant. | 0.0022467 (0.00267792)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 120 (Month 4) | 0.0015054 (0.00148462) | 0.0013500 (0.00002828) | 0.0000833 (0.00014434)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 360 (Month 12) | 0.0009971 (0.00173995) | 0.0000400 (NA) — SD was not estimable for a single participant. | 0.0003185 (0.00045043)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 15 | 0.0007662 (0.00172488) | 0.0030100 (0.00425678) | 0.0029133 (0.00493389)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0035320 (0.00412765) | 0.0050000 (0.00707107) | 0.0050000 (0.00866025)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0057832 (0.02013270) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 105 | 0.0037280 (0.00833606) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0063267 (0.01095811)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0017955 (0.00255443) | 0.0041500 (0.00586899) | 0.0049800 (0.00862561)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0025411 (0.00555028) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0480000 (0.02828427)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 15 | 0.0007143 (0.00197846) | 0.0010000 (0.00141421) | 0.0009033 (0.00156462)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1) | 0.0059520 (0.00996730) | 0.0145000 (0.02050610) | 0.0050000 (0.00500000)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3) | 0.0070000 (0.01086278) | 0.0060000 (0.00848528) | 0.0043333 (0.00585947)
  FNg-, IL2+, TNFa-, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  FNg-, IL2+, TNFa-, DENV-1, prME, Day 105 | 0.0046000 (0.00638749) | 0.0100000 (NA) — SD was not estimable for a single participant. | 0.0040000 (0.00608276)
  FNg-, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  FNg-, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4) | 0.0057273 (0.00553337) | 0.0000000 (0.00000000) | 0.0030000 (0.00519615)
  FNg-, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  FNg-, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12) | 0.0095556 (0.01255101) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0205000 (0.01060660)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 15 | 0.0098571 (0.02431930) | 0.0250000 (0.03535534) | 0.0376667 (0.01569501)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0063500 (0.01307177) | 0.0000000 (0.00000000) | 0.0466667 (0.08082904)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0040542 (0.01131730) | 0.0000000 (0.00000000) | 0.0310000 (0.04293018)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 105 | 0.0147960 (0.02254635) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0733333 (0.11846237)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0192727 (0.03854372) | 0.0400000 (0.05656854) | 0.0580000 (0.06009992)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0537778 (0.07350813) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 15 | 0.0156338 (0.01341318) | 0.0345000 (0.00070711) | 0.0156567 (0.01987399)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0122825 (0.01207005) | 0.0126170 (0.00213122) | 0.0140527 (0.01124558)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0069514 (0.00806641) | 0.0024950 (0.00133643) | 0.0038167 (0.00109573)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 105 | 0.0085950 (0.00881973) | 0.0080000 (NA) — SD was not estimable for a single participant. | 0.0026967 (0.00223813)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0114250 (0.00754569) | 0.0070200 (0.00021213) | 0.0055467 (0.00026764)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0113109 (0.00863169) | 0.0013000 (NA) — SD was not estimable for a single participant. | 0.0020875 (0.00290267)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 15 | 0.0055626 (0.00618103) | 0.0069450 (0.00426385) | 0.0016633 (0.00144057)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0037906 (0.00471970) | 0.0058220 (0.00022910) | 0.0065793 (0.00473908)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0024256 (0.00231885) | 0.0024550 (0.00338704) | 0.0020033 (0.00186162)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 105 | 0.0011180 (0.00155249) | 0.0029100 (NA) — SD was not estimable for a single participant. | 0.0021767 (0.00293742)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0018340 (0.00213001) | 0.0006150 (0.00086974) | 0.0039667 (0.00308171)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0016511 (0.00156732) | 0.0012900 (NA) — SD was not estimable for a single participant. | 0.0032340 (0.00314804)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 15 | 0.0195281 (0.01605864) | 0.0345000 (0.02757716) | 0.0396233 (0.02896264)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0129087 (0.01001686) | 0.0339320 (0.03984971) | 0.0194627 (0.01535958)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0074276 (0.00487590) | 0.0110000 (0.01555635) | 0.0150933 (0.00694661)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 105 | 0.0066833 (0.00676771) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0109133 (0.00335871)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0061417 (0.00294097) | 0.0113650 (0.01014698) | 0.0142633 (0.00845533)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0051673 (0.00437134) | 0.0000200 (NA) — SD was not estimable for a single participant. | 0.0063440 (0.00014991)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 15 | 0.0122905 (0.01136975) | 0.0166300 (0.01466539) | 0.0158833 (0.01526418)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0086183 (0.00744631) | 0.0184670 (0.02212254) | 0.0049393 (0.00441403)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0049071 (0.00312169) | 0.0030300 (0.00428507) | 0.0027600 (0.00079265)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 105 | 0.0013000 (0.00209346) | 0.0028600 (NA) — SD was not estimable for a single participant. | 0.0003333 (0.00057735)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.0017842 (0.00228371) | 0.0049750 (0.00504167) | 0.0037833 (0.00366041)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0029951 (0.00407349) | 0.0000500 (NA) — SD was not estimable for a single participant. | 0.0012250 (0.00173241)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 15 | 0.0184117 (0.02426237) | 0.0855000 (0.01202082) | 0.0023033 (0.00268712)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0253419 (0.03739564) | 0.0681170 (0.01978909) | 0.0055893 (0.00486565)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0180388 (0.01628354) | 0.0261400 (0.01677257) | 0.0015433 (0.00167828)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 105 | 0.0155460 (0.00736598) | 0.0304700 (NA) — SD was not estimable for a single participant. | 0.0010267 (0.00177824)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0255438 (0.02222056) | 0.0345400 (NA) — SD was not estimable for a single participant. | 0.0046400 (0.00643170)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0188425 (0.01749239) | 0.0208000 (NA) — SD was not estimable for a single participant. | 0.0046440 (0.00532593)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 15 | 0.0022795 (0.00242556) | 0.0097000 (0.00608112) | 0.0175233 (0.01552713)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0077111 (0.00670335) | 0.0215985 (0.03042186) | 0.0106660 (0.00795335)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0043389 (0.00329533) | 0.0075000 (0.01060660) | 0.0064033 (0.00380907)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 105 | 0.0026940 (0.00293657) | 0.0036000 (NA) — SD was not estimable for a single participant. | 0.0074700 (0.00868520)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0034200 (0.00296355) | 0.0049350 (0.00509824) | 0.0060967 (0.00653743)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0043200 (0.00603465) | 0.0000300 (NA) — SD was not estimable for a single participant. | 0.0012700 (0.00179605)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 15 | 0.0066462 (0.00792826) | 0.0084785 (0.01063701) | 0.0032200 (0.00404490)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 30 (Month 1) | 0.0088740 (0.01159933) | 0.0041720 (0.00065337) | 0.0030600 (0.00204404)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 90 (Month 3) | 0.0033060 (0.00441884) | 0.0017200 (0.00243245) | 0.0007633 (0.00085043)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 105 | 0.0079900 (0.01211394) | 0.0000390 (NA) — SD was not estimable for a single participant. | 0.0043500 (0.00284628)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4) | 0.0053583 (0.00565641) | 0.0013750 (0.00194454) | 0.0026010 (0.00178568)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12) | 0.0030009 (0.00444490) | 0.0025000 (NA) — SD was not estimable for a single participant. | 0.0008885 (0.00125653)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 15 | 0.0015118 (0.00191718) | 0.0015700 (0.00222032) | 0.0004667 (0.00080829)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1) | 0.0021769 (0.00268205) | 0.0047200 (0.00667509) | 0.0005833 (0.00101036)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3) | 0.0010054 (0.00138756) | 0.0000650 (0.00009192) | 0.0005967 (0.00103346)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 105 | 0.0016500 (0.00232157) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0005400 (0.00093531)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4) | 0.0006177 (0.00102890) | 0.0000000 (0.00000000) | 0.0008543 (0.00093306)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12) | 0.0006709 (0.00088977) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0010335 (0.00146159)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 15 | 0.0063455 (0.00700260) | 0.0061800 (0.00004243) | 0.0146700 (0.01675231)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 30 (Month 1) | 0.0099232 (0.01006738) | 0.0043520 (0.00203364) | 0.0085767 (0.00753694)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 90 (Month 3) | 0.0041648 (0.00370931) | 0.0016750 (0.00013435) | 0.0016000 (0.00277128)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 105 | 0.0062433 (0.00940730) | 0.0005200 (NA) — SD was not estimable for a single participant. | 0.0040567 (0.00418584)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4) | 0.0036216 (0.00439516) | 0.0012550 (0.00177484) | 0.0052677 (0.00341188)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12) | 0.0016830 (0.00264616) | 0.0012200 (NA) — SD was not estimable for a single participant. | 0.0016115 (0.00102601)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 15 | 0.0039528 (0.00428498) | 0.0011750 (0.00166170) | 0.0062000 (0.00507572)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 30 (Month 1) | 0.0043484 (0.00418555) | 0.0027520 (0.00121340) | 0.0020900 (0.00092677)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 90 (Month 3) | 0.0019436 (0.00233770) | 0.0007700 (0.00108894) | 0.0001920 (0.00033255)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 105 | 0.0012450 (0.00195501) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4) | 0.0014041 (0.00169202) | 0.0014300 (0.00202233) | 0.0001777 (0.00030773)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12) | 0.0009221 (0.00118263) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003085 (0.00043628)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 15 | 0.0063457 (0.00739280) | 0.0276900 (0.03013689) | 0.0023867 (0.00266356)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1) | 0.0136346 (0.01827227) | 0.0124520 (0.00519299) | 0.0025633 (0.00102627)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3) | 0.0102555 (0.00890732) | 0.0107550 (0.00034648) | 0.0009733 (0.00168586)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 105 | 0.0086980 (0.00422567) | 0.0081900 (NA) — SD was not estimable for a single participant. | 0.0015767 (0.00273087)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4) | 0.0096186 (0.00919641) | 0.0014200 (NA) — SD was not estimable for a single participant. | 0.0006143 (0.00065878)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12) | 0.0051619 (0.00721208) | 0.0130000 (NA) — SD was not estimable for a single participant. | 0.0013275 (0.00066397)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 15 | 0.0012506 (0.00145149) | 0.0034600 (0.00052326) | 0.0049867 (0.00557140)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1) | 0.0041405 (0.00370046) | 0.0030320 (0.00143967) | 0.0044700 (0.00201167)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3) | 0.0023277 (0.00290426) | 0.0029050 (0.00410829) | 0.0034137 (0.00278951)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 105 | 0.0025060 (0.00269757) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0020167 (0.00116453)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4) | 0.0019454 (0.00182333) | 0.0014450 (0.00204354) | 0.0012343 (0.00133427)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12) | 0.0007733 (0.00127164) | 0.0012300 (NA) — SD was not estimable for a single participant. | 0.0004275 (0.00058336)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 15 | 0.0060766 (0.00449815) | 0.0428850 (0.01611496) | 0.0240633 (0.03025849)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0037728 (0.00410557) | 0.0185620 (0.01051892) | 0.0079800 (0.00575490)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0015660 (0.00222761) | 0.0032600 (0.00217789) | 0.0057033 (0.00286514)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 105 | 0.0043250 (0.00738836) | 0.0045900 (NA) — SD was not estimable for a single participant. | 0.0056000 (0.00592666)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0046358 (0.00481391) | 0.0035500 (0.00308299) | 0.0027843 (0.00263947)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0039912 (0.00426930) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0016035 (0.00145169)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 15 | 0.0020367 (0.00200211) | 0.0119550 (0.01460176) | 0.0034600 (0.00072547)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0009933 (0.00141721) | 0.0047720 (0.00660155) | 0.0009560 (0.00076228)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0005400 (0.00102516) | 0.0018050 (0.00255266) | 0.0002240 (0.00038798)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 105 | 0.0026620 (0.00525083) | 0.0000430 (NA) — SD was not estimable for a single participant. | 0.0018267 (0.00165908)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0005960 (0.00082714) | 0.0006150 (0.00086974) | 0.0015343 (0.00028065)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0009544 (0.00127228) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0010335 (0.00146159)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 15 | 0.0090109 (0.00856650) | 0.0543850 (0.05359162) | 0.0473333 (0.03165965)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0064879 (0.00601416) | 0.0269820 (0.03538079) | 0.0190567 (0.01080034)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0026280 (0.00337824) | 0.0067600 (0.00956008) | 0.0078667 (0.00525903)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 105 | 0.0031033 (0.00107483) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0076500 (0.00526430)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0028733 (0.00244337) | 0.0062700 (0.00886712) | 0.0048743 (0.00332532)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0019966 (0.00189583) | 0.0000200 (NA) — SD was not estimable for a single participant. | 0.0022035 (0.00064559)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 15 | 0.0063809 (0.00759632) | 0.0236700 (0.03338958) | 0.0097900 (0.01084422)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0031547 (0.00278886) | 0.0170245 (0.02400698) | 0.0018733 (0.00038760)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0013470 (0.00190419) | 0.0007900 (0.00111723) | 0.0001920 (0.00033255)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 105 | 0.0014450 (0.00172311) | 0.0017300 (NA) — SD was not estimable for a single participant. | 0.0013200 (0.00117235)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.0009200 (0.00124907) | 0.0062700 (0.00886712) | 0.0031343 (0.00307798)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0032012 (0.00384132) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003085 (0.00043628)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 15 | 0.0043954 (0.00510405) | 0.0878850 (0.01328654) | 0.0024367 (0.00211519)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0079454 (0.00902785) | 0.0505620 (0.00486207) | 0.0035200 (0.00305210)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0054914 (0.00581130) | 0.0224000 (0.00582656) | 0.0014500 (0.00146010)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 105 | 0.0114020 (0.01790945) | 0.0284700 (NA) — SD was not estimable for a single participant. | 0.0016133 (0.00163026)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0070050 (0.00365273) | 0.0165400 (NA) — SD was not estimable for a single participant. | 0.0032910 (0.00127837)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0065866 (0.00631099) | 0.0188000 (NA) — SD was not estimable for a single participant. | 0.0022325 (0.00194384)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 15 | 0.0024265 (0.00372846) | 0.0270400 (0.03710896) | 0.0520867 (0.05471529)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0045850 (0.00682112) | 0.0245000 (0.03464823) | 0.0250400 (0.03055440)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0015112 (0.00306508) | 0.0077600 (0.01097430) | 0.0107867 (0.01190998)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 105 | 0.0011860 (0.00163110) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0098533 (0.00613096)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0013082 (0.00189986) | 0.0134350 (0.01711906) | 0.0126110 (0.01695829)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0036009 (0.00879474) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0004275 (0.00058336)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 15 | 0.0075520 (0.00844484) | 0.0330950 (0.02107885) | 0.0096033 (0.00523661)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 30 (Month 1) | 0.0080525 (0.01055229) | 0.0055700 (0.00255973) | 0.0057660 (0.00370940)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 90 (Month 3) | 0.0034662 (0.00388476) | 0.0030950 (0.00437699) | 0.0020620 (0.00178653)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 105 | 0.0063400 (0.00932154) | 0.0017500 (NA) — SD was not estimable for a single participant. | 0.0036733 (0.00290569)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 120 (Month 4) | 0.0051208 (0.00397179) | 0.0021100 (0.00104652) | 0.0010100 (0.00156272)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 360 (Month 12) | 0.0024600 (0.00277472) | 0.0013000 (NA) — SD was not estimable for a single participant. | 0.0029585 (0.00170908)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 15 | 0.0020206 (0.00260390) | 0.0042250 (0.00290621) | 0.0026533 (0.00089891)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 30 (Month 1) | 0.0020286 (0.00206735) | 0.0000000 (0.00000000) | 0.0014793 (0.00041333)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 90 (Month 3) | 0.0009626 (0.00123421) | 0.0016200 (0.00229103) | 0.0013687 (0.00170601)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 105 | 0.0003300 (0.00056303) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0005433 (0.00094108)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 120 (Month 4) | 0.0004290 (0.00077370) | 0.0000000 (0.00000000) | 0.0004800 (0.00083138)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 360 (Month 12) | 0.0009997 (0.00125950) | 0.0000400 (NA) — SD was not estimable for a single participant. | 0.0003635 (0.00051407)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 15 | 0.0101574 (0.01135027) | 0.0455950 (0.00084146) | 0.0346667 (0.01833939)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 30 (Month 1) | 0.0079673 (0.00830325) | 0.0056000 (0.00637810) | 0.0117927 (0.00809815)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 90 (Month 3) | 0.0039573 (0.00329832) | 0.0031250 (0.00427800) | 0.0057620 (0.00888965)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 105 | 0.0045767 (0.00294576) | 0.0005200 (NA) — SD was not estimable for a single participant. | 0.0025567 (0.00157912)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 120 (Month 4) | 0.0035933 (0.00301672) | 0.0031800 (0.00055154) | 0.0034733 (0.00388177)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 360 (Month 12) | 0.0016788 (0.00208657) | 0.0012300 (NA) — SD was not estimable for a single participant. | 0.0029385 (0.00085065)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 15 | 0.0044780 (0.00694930) | 0.0130950 (0.00154856) | 0.0065773 (0.00619340)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 30 (Month 1) | 0.0044494 (0.00362591) | 0.0060550 (0.00856306) | 0.0013160 (0.00044863)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 90 (Month 3) | 0.0022088 (0.00270445) | 0.0037850 (0.00535280) | 0.0002120 (0.00036719)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 105 | 0.0006333 (0.00098508) | 0.0011700 (NA) — SD was not estimable for a single participant. | 0.0005267 (0.00091221)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 120 (Month 4) | 0.0015674 (0.00117213) | 0.0000000 (0.00000000) | 0.0011733 (0.00203227)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 360 (Month 12) | 0.0006924 (0.00099937) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0004310 (0.00060953)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 15 | 0.0066937 (0.00722100) | 0.0915950 (0.08259714) | 0.0062000 (0.00563205)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 30 (Month 1) | 0.0079714 (0.00798185) | 0.0441800 (0.02979748) | 0.0015410 (0.00085791)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 90 (Month 3) | 0.0074104 (0.00838499) | 0.0197800 (0.01241680) | 0.0011100 (0.00192258)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 105 | 0.0086560 (0.01075630) | 0.0087000 (NA) — SD was not estimable for a single participant. | 0.0010400 (0.00180133)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 120 (Month 4) | 0.0060286 (0.00431794) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003600 (0.00062354)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 360 (Month 12) | 0.0032638 (0.00481301) | 0.0138000 (NA) — SD was not estimable for a single participant. | 0.0005985 (0.00084641)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 15 | 0.0019264 (0.00178363) | 0.0039900 (0.00127279) | 0.0442107 (0.04821126)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 30 (Month 1) | 0.0044725 (0.00358891) | 0.0075900 (0.00639225) | 0.0092893 (0.00950700)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 90 (Month 3) | 0.0014555 (0.00277488) | 0.0029200 (0.00412950) | 0.0020720 (0.00091517)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 105 | 0.0019320 (0.00391432) | 0.0006500 (NA) — SD was not estimable for a single participant. | 0.0022200 (0.00384515)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 120 (Month 4) | 0.0018336 (0.00149423) | 0.0006650 (0.00094045) | 0.0021167 (0.00171704)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 360 (Month 12) | 0.0007334 (0.00095378) | 0.0000300 (NA) — SD was not estimable for a single participant. | 0.0004200 (0.00059397)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 15 | 0.0024433 (0.00478745) | 0.0000000 (0.00000000) | 0.0064967 (0.00809850)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0087252 (0.01274292) | 0.0000000 (0.00000000) | 0.0004767 (0.00082561)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0022710 (0.00378206) | 0.0000000 (0.00000000) | 0.0303333 (0.05253887)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 105 | 0.0032733 (0.00561714) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0096600 (0.01002032)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0054000 (0.00546757) | 0.0014550 (0.00205768) | 0.0101467 (0.01719490)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0057482 (0.01145463) | 0.0010000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 15 | 0.0023484 (0.00373999) | 0.0000000 (0.00000000) | 0.0019433 (0.00336595)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0027084 (0.00347026) | 0.0115000 (0.00636396) | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0004250 (0.00128026) | 0.0000000 (0.00000000) | 0.0060000 (0.01039230)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 105 | 0.0034460 (0.00473493) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003333 (0.00057735)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0040230 (0.00533216) | 0.0051500 (0.00728320) | 0.0026467 (0.00458416)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0028144 (0.00395317) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0175000 (0.00070711)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 15 | 0.0020638 (0.00335443) | 0.0000000 (0.00000000) | 0.0045367 (0.00785774)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0061967 (0.01073863) | 0.0030000 (0.00424264) | 0.0050000 (0.00866025)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0028243 (0.00657932) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 105 | 0.0043583 (0.00586855) | 0.0010000 (NA) — SD was not estimable for a single participant. | 0.0016667 (0.00152753)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0041158 (0.00481914) | 0.0056500 (0.00799031) | 0.0109800 (0.00962191)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0043409 (0.00775431) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 15 | 0.0029114 (0.00457042) | 0.0040100 (0.00567100) | 0.0095367 (0.01244163)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0060424 (0.00716413) | 0.0000000 (0.00000000) | 0.0081633 (0.00851998)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0029867 (0.00872447) | 0.0025000 (0.00353553) | 0.0134067 (0.02049576)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 105 | 0.0023333 (0.00297921) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.0031367 (0.00432011) | 0.0015750 (0.00222739) | 0.0053133 (0.00920296)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0074518 (0.01318948) | 0.0010000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 15 | 0.0077311 (0.01847127) | 0.0080100 (0.00425678) | 0.0044800 (0.00577678)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0105571 (0.00966628) | 0.0120000 (0.00989949) | 0.0074967 (0.00705266)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0085371 (0.01020675) | 0.0090000 (0.00282843) | 0.0017500 (0.00303109)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 105 | 0.0227280 (0.03716463) | 0.0050000 (NA) — SD was not estimable for a single participant. | 0.0069933 (0.00607619)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0100288 (0.01429998) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0099800 (0.01728587)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0138388 (0.01736932) | 0.0020000 (NA) — SD was not estimable for a single participant. | 0.0485000 (0.03181981)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 15 | 0.0006881 (0.00163780) | 0.0000000 (0.00000000) | 0.0222033 (0.03371578)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0083430 (0.01049993) | 0.0000000 (0.00000000) | 0.0081633 (0.00851998)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0039411 (0.00506722) | 0.0075000 (0.01060660) | 0.0193333 (0.03348632)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 105 | 0.0057280 (0.00796431) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0019900 (0.00262874)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0058000 (0.00727803) | 0.0031500 (0.00445477) | 0.0023100 (0.00400104)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0055411 (0.00703655) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0770000 (0.00989949)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 15 | 0.0048771 (0.00581334) | 0.0010000 (0.00141421) | 0.0055700 (0.00649882)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 30 (Month 1) | 0.0110019 (0.01406371) | 0.0010000 (0.00141421) | 0.0033333 (0.00577350)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 90 (Month 3) | 0.0048095 (0.00757376) | 0.0055000 (0.00212132) | 0.0146667 (0.01616581)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 105 | 0.0066667 (0.01114750) | 0.0090000 (NA) — SD was not estimable for a single participant. | 0.0086667 (0.01078579)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4) | 0.0131667 (0.01259750) | 0.0000000 (0.00000000) | 0.0056667 (0.00550757)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12) | 0.0045455 (0.00706206) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0025000 (0.00353553)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 15 | 0.0027368 (0.00646222) | 0.0005000 (0.00070711) | 0.0032367 (0.00302788)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1) | 0.0042653 (0.00817199) | 0.0190000 (0.02687006) | 0.0066667 (0.01154701)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3) | 0.0041111 (0.00669406) | 0.0050000 (0.00707107) | 0.0173333 (0.02746513)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 105 | 0.0008000 (0.00130384) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4) | 0.0092000 (0.01536808) | 0.0000000 (0.00000000) | 0.0080000 (0.00608276)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12) | 0.0115556 (0.01326755) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0340000 (0.02404163)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 15 | 0.0019248 (0.00358174) | 0.0030000 (0.00424264) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 30 (Month 1) | 0.0051448 (0.00695615) | 0.0000000 (0.00000000) | 0.0130000 (0.00556776)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 90 (Month 3) | 0.0054286 (0.00796600) | 0.0035000 (0.00494975) | 0.0043333 (0.00585947)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 105 | 0.0021667 (0.00325064) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0016667 (0.00288675)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4) | 0.0079167 (0.00674818) | 0.0000000 (0.00000000) | 0.0116667 (0.01386843)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12) | 0.0058182 (0.00726386) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0040000 (0.00565685)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 15 | 0.0029248 (0.00608645) | 0.0030000 (0.00424264) | 0.0082367 (0.01120795)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 30 (Month 1) | 0.0050019 (0.00532053) | 0.0015000 (0.00212132) | 0.0030000 (0.00300000)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 90 (Month 3) | 0.0040476 (0.00569628) | 0.0080000 (0.01131371) | 0.0063333 (0.00709460)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 105 | 0.0020000 (0.00400000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4) | 0.0040000 (0.00645262) | 0.0000000 (0.00000000) | 0.0003333 (0.00057735)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12) | 0.0063636 (0.00868646) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0155000 (0.02192031)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 15 | 0.0033889 (0.00726101) | 0.0010000 (0.00141421) | 0.0140067 (0.02424294)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1) | 0.0105906 (0.01290502) | 0.0075000 (0.01060660) | 0.0056667 (0.00513160)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3) | 0.0081765 (0.01052518) | 0.0225000 (0.00494975) | 0.0100000 (0.00916515)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 105 | 0.0106000 (0.01436315) | 0.0270000 (NA) — SD was not estimable for a single participant. | 0.0026667 (0.00461880)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4) | 0.0138750 (0.01167950) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0116667 (0.00776745)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12) | 0.0388750 (0.04258584) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0360000 (0.01272792)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 15 | 0.0018571 (0.00381164) | 0.0005000 (0.00070711) | 0.0094100 (0.01524580)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1) | 0.0100520 (0.00984572) | 0.0000000 (0.00000000) | 0.0060000 (0.00519615)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3) | 0.0052105 (0.00611536) | 0.0050000 (0.00707107) | 0.0113333 (0.01962991)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 105 | 0.0048000 (0.00672309) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4) | 0.0063636 (0.00569689) | 0.0000000 (0.00000000) | 0.0026667 (0.00461880)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12) | 0.0035556 (0.00538774) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0595000 (0.01343503)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 15 | 0.0007143 (0.00327327) | 0.0000000 (0.00000000) | 0.0210000 (0.03637307)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0033810 (0.00696043) | 0.0000000 (0.00000000) | 0.0233333 (0.04041452)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0038586 (0.01248055) | 0.0000000 (0.00000000) | 0.0100000 (0.01732051)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 105 | 0.0009967 (0.00199200) | 0.0200000 (NA) — SD was not estimable for a single participant. | 0.0133333 (0.02309401)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0070000 (0.01205291) | 0.0000000 (0.00000000) | 0.0053333 (0.00923760)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0233636 (0.04872838) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0050000 (0.00707107)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 15 | 0.0330526 (0.05651693) | 0.0450000 (0.06363961) | 0.0976667 (0.05173329)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0089474 (0.01355021) | 0.0000000 (0.00000000) | 0.1373333 (0.08247020)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0102239 (0.02008526) | 0.0600000 (0.08485281) | 0.0596667 (0.06961561)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 105 | 0.0501960 (0.10057640) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.1293333 (0.19110556)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0088000 (0.01360392) | 0.0050000 (0.00707107) | 0.0413333 (0.04006661)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0466667 (0.05889822) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0050000 (0.00707107)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 15 | 0.0020952 (0.00545807) | 0.0000000 (0.00000000) | 0.0176667 (0.01078579)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0015714 (0.00413003) | 0.0000000 (0.00000000) | 0.0500000 (0.07000000)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0060967 (0.01538351) | 0.0050000 (0.00707107) | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 105 | 0.0031633 (0.00681587) | 0.0400000 (NA) — SD was not estimable for a single participant. | 0.0466667 (0.07234178)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0064167 (0.01195034) | 0.0200000 (0.02828427) | 0.0020000 (0.00346410)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0322727 (0.05355388) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 15 | 0.0030952 (0.00770652) | 0.0850000 (0.12020815) | 0.0710000 (0.05179768)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0025714 (0.00517273) | 0.0100000 (0.01414214) | 0.0996667 (0.11571661)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0025252 (0.00822553) | 0.0300000 (0.04242641) | 0.0336667 (0.04147690)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 105 | 0.0031633 (0.00567028) | 0.0100000 (NA) — SD was not estimable for a single participant. | 0.0700000 (0.12124356)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.0063333 (0.00867948) | 0.0250000 (0.03535534) | 0.0846667 (0.10346658)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0237273 (0.04557212) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 15 | 0.0109444 (0.02263644) | 0.0450000 (0.06363961) | 0.1443333 (0.09152231)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0254118 (0.05545388) | 0.0850000 (0.12020815) | 0.1506667 (0.07759725)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0341782 (0.05499065) | 0.0500000 (0.07071068) | 0.0906667 (0.05138417)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 105 | 0.1933960 (0.34758253) | 0.0200000 (NA) — SD was not estimable for a single participant. | 0.1556667 (0.14424401)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0088750 (0.01786807) | 0.0200000 (NA) — SD was not estimable for a single participant. | 0.1313333 (0.16341767)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0786250 (0.07674250) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0350000 (0.02121320)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 15 | 0.0007143 (0.00327327) | 0.0200000 (0.02828427) | 0.0500000 (0.07810250)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0050500 (0.01240745) | 0.0000000 (0.00000000) | 0.0570000 (0.06408588)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0116332 (0.02395900) | 0.0450000 (0.06363961) | 0.0133333 (0.02309401)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 105 | 0.0049960 (0.01117140) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0500000 (0.07000000)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0040909 (0.00870005) | 0.0200000 (0.02828427) | 0.0346667 (0.03500476)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0546667 (0.07867655) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 15 | 0.0045624 (0.00373863) | 0.0132800 (0.01657458) | 0.0156033 (0.01522844)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0037701 (0.00361243) | 0.0224970 (0.02915118) | 0.0166927 (0.02121306)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0019732 (0.00203413) | 0.0073800 (0.00794788) | 0.0066433 (0.00434298)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 105 | 0.0010780 (0.00144028) | 0.0005900 (NA) — SD was not estimable for a single participant. | 0.0065467 (0.00607425)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0029255 (0.00304491) | 0.0072700 (0.01028133) | 0.0087367 (0.01165157)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0024944 (0.00265027) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0065440 (0.00147927)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 15 | 0.0020067 (0.00349245) | 0.0017650 (0.00249609) | 0.0027067 (0.00204500)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1) | 0.0027715 (0.00491943) | 0.0084820 (0.01063206) | 0.0062267 (0.00469696)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3) | 0.0009887 (0.00117522) | 0.0008700 (0.00123037) | 0.0009033 (0.00078932)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 105 | 0.0011940 (0.00117362) | 0.0000290 (NA) — SD was not estimable for a single participant. | 0.0009600 (0.00088386)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4) | 0.0020154 (0.00212428) | 0.0013950 (0.00007778) | 0.0016910 (0.00108924)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12) | 0.0004596 (0.00090723) | 0.0012300 (NA) — SD was not estimable for a single participant. | 0.0009050 (0.00127986)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 15 | 0.0029003 (0.00272483) | 0.0194500 (0.02521543) | 0.0487733 (0.04944810)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0013431 (0.00157750) | 0.0154820 (0.02053155) | 0.0255367 (0.02610415)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0009037 (0.00153323) | 0.0057600 (0.00814587) | 0.0140600 (0.01672199)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 105 | 0.0024900 (0.00217522) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0164733 (0.01680245)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0007918 (0.00151918) | 0.0057700 (0.00816001) | 0.0145877 (0.01618069)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0014281 (0.00135883) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0019985 (0.00102036)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 15 | 0.0023851 (0.00349970) | 0.0054855 (0.00665317) | 0.0347667 (0.03185692)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 30 (Month 1) | 0.0019231 (0.00285971) | 0.0025200 (0.00213546) | 0.0119560 (0.00976035)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 90 (Month 3) | 0.0012856 (0.00145620) | 0.0023950 (0.00338704) | 0.0028307 (0.00290989)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 105 | 0.0004400 (0.00061192) | 0.0005900 (NA) — SD was not estimable for a single participant. | 0.0047467 (0.00638064)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 120 (Month 4) | 0.0020605 (0.00152830) | 0.0021700 (0.00306884) | 0.0043733 (0.00330736)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 360 (Month 12) | 0.0007457 (0.00106006) | 0.0000300 (NA) — SD was not estimable for a single participant. | 0.0009135 (0.00126784)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 15 | 0.0006690 (0.00177413) | 0.0000000 (0.00000000) | 0.0182233 (0.01991388)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0037725 (0.00540746) | 0.0000000 (0.00000000) | 0.0034967 (0.00303810)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0016332 (0.00284966) | 0.0000000 (0.00000000) | 0.0176733 (0.02887941)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 105 | 0.0024340 (0.00417459) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0038967 (0.00400400)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0026618 (0.00395446) | 0.0006850 (0.00096874) | 0.0020133 (0.00348720)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0042078 (0.00647931) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0170000 (0.02404163)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 15 | 0.0026390 (0.00478957) | 0.0030000 (0.00424264) | 0.0126667 (0.02193931)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1) | 0.0052020 (0.00685207) | 0.0085000 (0.01202082) | 0.0060000 (0.00871780)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3) | 0.0022105 (0.00432793) | 0.0000000 (0.00000000) | 0.0173333 (0.03002221)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 105 | 0.0040000 (0.00616441) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0013333 (0.00230940)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4) | 0.0047273 (0.00864975) | 0.0000000 (0.00000000) | 0.0113333 (0.01001665)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12) | 0.0103333 (0.01298075) | 0.0020000 (NA) — SD was not estimable for a single participant. | 0.0200000 (0.01272792)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 15 | 0.0064286 (0.01567345) | 0.0300000 (0.04242641) | 0.0476667 (0.06368935)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0037000 (0.00877856) | 0.0000000 (0.00000000) | 0.0700000 (0.10440307)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0040016 (0.01133985) | 0.0150000 (0.02121320) | 0.0370000 (0.03517101)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 105 | 0.0123960 (0.01897351) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0433333 (0.07505553)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0055455 (0.00831100) | 0.0200000 (0.02828427) | 0.0580000 (0.05031898)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0488889 (0.08153595) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0250000 (0.03535534)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 15 | 0.0042128 (0.00495148) | 0.0280000 (0.01272792) | 0.0013133 (0.00119605)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0041551 (0.00511084) | 0.0273970 (0.03353525) | 0.0045693 (0.00367278)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0018916 (0.00291470) | 0.0120550 (0.01689278) | 0.0010800 (0.00183608)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 105 | 0.0007540 (0.00168600) | 0.0064500 (NA) — SD was not estimable for a single participant. | 0.0004667 (0.00080829)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0028073 (0.00241349) | 0.0101050 (0.01051468) | 0.0018300 (0.00189834)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0034077 (0.00388535) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0009250 (0.00130815)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 15 | 0.0010586 (0.00123430) | 0.0072000 (0.00026870) | 0.0002150 (0.00037239)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1) | 0.0015226 (0.00145884) | 0.0106670 (0.00471357) | 0.0004867 (0.00084293)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3) | 0.0013921 (0.00146570) | 0.0009150 (0.00129401) | 0.0002013 (0.00034872)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 105 | 0.0020120 (0.00343865) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0012300 (0.00111665)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4) | 0.0016538 (0.00147798) | 0.0013500 (0.00002828) | 0.0010277 (0.00133012)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12) | 0.0005131 (0.00105742) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000010 (0.00000141)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 15 | 0.0019679 (0.00226430) | 0.0298850 (0.02884289) | 0.0026567 (0.00243097)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0014351 (0.00201558) | 0.0349770 (0.04811579) | 0.0028800 (0.00258519)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0005243 (0.00078972) | 0.0102600 (0.01450983) | 0.0006033 (0.00104500)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 105 | 0.0021520 (0.00374127) | 0.0012200 (NA) — SD was not estimable for a single participant. | 0.0014633 (0.00168138)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0010900 (0.00094653) | 0.0082700 (0.01169555) | 0.0021233 (0.00266215)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0009091 (0.00135131) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003085 (0.00043628)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 15 | 0.0021766 (0.00325195) | 0.0180950 (0.00296278) | 0.0010083 (0.00123090)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 30 (Month 1) | 0.0019537 (0.00217059) | 0.0150950 (0.02123442) | 0.0018260 (0.00126872)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 90 (Month 3) | 0.0011930 (0.00181994) | 0.0050000 (0.00707107) | 0.0021353 (0.00311525)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 105 | 0.0013140 (0.00138036) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0015733 (0.00166677)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 120 (Month 4) | 0.0009293 (0.00129407) | 0.0019950 (0.00094045) | 0.0006533 (0.00106308)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 360 (Month 12) | 0.0006534 (0.00095082) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000010 (0.00000141)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 15 | 0.0010538 (0.00210085) | 0.0035100 (0.00352139) | 0.0018700 (0.00323894)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0053990 (0.00689308) | 0.0010000 (0.00141421) | 0.0051633 (0.00690000)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0027358 (0.00322179) | 0.0010000 (0.00141421) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 105 | 0.0014640 (0.00259932) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0043267 (0.00749401)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0057182 (0.00781389) | 0.0013200 (0.00186676) | 0.0043133 (0.00447823)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0034000 (0.00501189) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0120000 (0.01697056)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 15 | 0.0048771 (0.00855424) | 0.0030000 (0.00282843) | 0.0032367 (0.00336125)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1) | 0.0055520 (0.00738344) | 0.0030000 (0.00424264) | 0.0073333 (0.01021437)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3) | 0.0032105 (0.00491685) | 0.0060000 (0.00141421) | 0.0070000 (0.01212436)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 105 | 0.0006000 (0.00134164) | 0.0100000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4) | 0.0093636 (0.01344078) | 0.0000000 (0.00000000) | 0.0040000 (0.00692820)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12) | 0.0072222 (0.01328324) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0145000 (0.02050610)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 15 | 0.0128095 (0.02841939) | 0.1150000 (0.16263456) | 0.1576667 (0.05173329)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0137000 (0.02625202) | 0.0250000 (0.03535534) | 0.1056667 (0.10390541)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0117384 (0.01908793) | 0.0750000 (0.10606602) | 0.0540000 (0.03751000)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 105 | 0.0123960 (0.01978191) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0733333 (0.08736895)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0190000 (0.02560078) | 0.0400000 (0.05656854) | 0.0880000 (0.07830709)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0607778 (0.06849777) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0600000 (0.08485281)

14. Secondary Outcome: Phenotype Characterization of Cellular Immune Response to TDV Assessed as Percentage of Total CD8+ T Cells by Intracellular Cytokine Staining (ICS)
Description: Phenotype characterization of cellular immune response was performed in a subset of participants with IFN- γ ELISPOT responses >50 SFC/10^6 cells and availability of sufficient cells. Markers included CD4, CD8, IFN-γ, tumor necrosis factor-alpha (TNF-α) and interleukin-2 (IL-2). The peptide pools included C, NS1, NS2/4, NS3, NS5 for DENV-2 and prME for DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: Days 15, 30 (Month 1), 90 (Month 3), 105, 120 (Month 4), and 360 (Month 12)
Population: ICS Subset included participants from PPS (all participants in the FAS who had no major protocol violations) who had IFN-γ ELISPOT responses >50 SFC/10^6 PBMCs and availability of sufficient cells for analysis. Number analyzed is the number of participants with data available for analysis for the specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of CD8+ T cells
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive
Number analyzed (Participants) | 21 | 2 | 3
percentage of CD8+ T cells
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 15 | 0.0056604 (0.01627332) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0047007 (0.01502896) | 0.0000750 (0.00010607) | 0.0008833 (0.00152998)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0014703 (0.00267161) | 0.0026650 (0.00376888) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 105 | 0.0000000 (0.00000000) | 0.0013600 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0082836 (0.01892632) | 0.0008700 (0.00123037) | 0.0009333 (0.00161658)
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0016900 (0.00330848) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 15 | 0.0024200 (0.00800006) | 0.0000000 (0.00000000) | 0.0025900 (0.00448601)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1) | 0.0055525 (0.02087829) | 0.0000000 (0.00000000) | 0.0003040 (0.00052654)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3) | 0.0011563 (0.00285872) | 0.0000000 (0.00000000) | 0.0009200 (0.00159349)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 105 | 0.0014160 (0.00316627) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0004400 (0.00076210)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4) | 0.0039800 (0.01170301) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12) | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 15 | 0.0144803 (0.02730440) | 0.0025450 (0.00359917) | 0.0023033 (0.00203952)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0370610 (0.11025384) | 0.0332550 (0.03782314) | 0.0102833 (0.01232115)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0241643 (0.03587491) | 0.0205000 (0.02899138) | 0.0075367 (0.01031316)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 105 | 0.0077060 (0.00514342) | 0.0013600 (NA) — SD was not estimable for a single participant. | 0.0043933 (0.00382467)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0602155 (0.15407711) | 0.0198650 (0.02809335) | 0.0059600 (0.00785521)
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0112811 (0.01654078) | 0.0031000 (NA) — SD was not estimable for a single participant. | 0.0021250 (0.00300520)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 15 | 0.0159699 (0.04359877) | 0.0017000 (0.00240416) | 0.0004900 (0.00084870)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 30 (Month 1) | 0.0707734 (0.25211961) | 0.0278700 (0.01820093) | 0.0029790 (0.00433441)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 90 (Month 3) | 0.0288527 (0.08127031) | 0.0117600 (0.01066317) | 0.0032033 (0.00444653)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 105 | 0.0070820 (0.01452614) | 0.0040800 (NA) — SD was not estimable for a single participant. | 0.0012633 (0.00114718)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 120 (Month 4) | 0.0560967 (0.15418829) | 0.0060000 (0.00848528) | 0.0022283 (0.00320135)
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-1, prME, Day 360 (Month 12) | 0.0019478 (0.00186916) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 15 | 0.0003281 (0.00087119) | 0.0008500 (0.00120208) | 0.0016667 (0.00288675)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0014660 (0.00368403) | 0.0070000 (0.00989949) | 0.0015217 (0.00263560)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0018853 (0.00779198) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 105 | 0.0008120 (0.00181569) | 0.0018800 (NA) — SD was not estimable for a single participant. | 0.0038700 (0.00670304)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0004069 (0.00077459) | 0.0000000 (0.00000000) | 0.0120000 (0.02078461)
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0017656 (0.00266025) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0312150 (0.02010305)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 15 | 0.0030481 (0.00520443) | 0.0000000 (0.00000000) | 0.0043333 (0.00378594)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 30 (Month 1) | 0.0029060 (0.00436453) | 0.0000000 (0.00000000) | 0.0023333 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 90 (Month 3) | 0.0040816 (0.00613449) | 0.0085000 (0.01202082) | 0.0023333 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 105 | 0.0000000 (0.00000000) | 0.0110000 (NA) — SD was not estimable for a single participant. | 0.0033333 (0.00305505)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 120 (Month 4) | 0.0020000 (0.00300000) | 0.0000000 (0.00000000) | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-1, prME, Day 360 (Month 12) | 0.0062678 (0.01052641) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0070000 (0.00848528)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 15 | 0.0148095 (0.02511227) | 0.0195000 (0.01767767) | 0.0060000 (0.01039230)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 30 (Month 1) | 0.0115435 (0.01646364) | 0.0235000 (0.01343503) | 0.0253333 (0.03106981)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 90 (Month 3) | 0.0093311 (0.01492871) | 0.0250000 (0.03535534) | 0.0316667 (0.03102150)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 105 | 0.0246000 (0.02815670) | 0.0110000 (NA) — SD was not estimable for a single participant. | 0.0266667 (0.04532475)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 120 (Month 4) | 0.0250255 (0.03675944) | 0.0295000 (0.03323402) | 0.0080000 (0.01385641)
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-1, prME, Day 360 (Month 12) | 0.0386067 (0.03656897) | 0.0030000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 15 | 0.0042606 (0.00562943) | 0.0025550 (0.00361332) | 0.0019520 (0.00148274)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0194350 (0.06157246) | 0.0088700 (0.01254407) | 0.0116087 (0.01939586)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0105474 (0.02561865) | 0.0055000 (0.00777817) | 0.0080000 (0.01385641)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 105 | 0.0006717 (0.00164524) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0016067 (0.00278283)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0090928 (0.01602139) | 0.0000000 (0.00000000) | 0.0134433 (0.02214271)
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0115891 (0.01525538) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003415 (0.00048295)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 15 | 0.0115911 (0.02556364) | 0.0034050 (0.00481540) | 0.0230000 (0.02523886)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0331987 (0.06119374) | 0.0022800 (0.00322441) | 0.0284400 (0.02579343)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0235620 (0.03383365) | 0.0034850 (0.00492853) | 0.0246667 (0.02247962)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 105 | 0.0246240 (0.03733209) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0220000 (0.02029778)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0097230 (0.01765134) | 0.0025150 (0.00355675) | 0.0270000 (0.03044667)
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0127111 (0.01056931) | 0.0030800 (NA) — SD was not estimable for a single participant. | 0.0370000 (0.05232590)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 15 | 0.0173215 (0.02522769) | 0.0258900 (0.03126826) | 0.0195800 (0.02908452)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0598512 (0.09417635) | 0.1423700 (0.17729995) | 0.0307000 (0.04702863)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0582231 (0.09890918) | 0.0672150 (0.08879140) | 0.0477333 (0.07132611)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 105 | 0.0113983 (0.01184397) | 0.0036900 (NA) — SD was not estimable for a single participant. | 0.0410800 (0.06836592)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0652592 (0.11485350) | 0.0815250 (0.11098041) | 0.0249567 (0.03147802)
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0482255 (0.06448748) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0038600 (0.00397394)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 15 | 0.0188293 (0.02998412) | 0.0054950 (0.00047376) | 0.0023870 (0.00145326)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0944508 (0.21411201) | 0.0699200 (0.09591196) | 0.0180433 (0.02775222)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0866393 (0.13212126) | 0.0516100 (0.06701958) | 0.0104300 (0.01696039)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 105 | 0.0439383 (0.05779160) | 0.0039700 (NA) — SD was not estimable for a single participant. | 0.0182000 (0.03014830)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.1042408 (0.16997426) | 0.0430000 (0.06081118) | 0.0129300 (0.01662924)
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0624582 (0.07686613) | 0.0062300 (NA) — SD was not estimable for a single participant. | 0.0005050 (0.00071418)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 15 | 0.0008767 (0.00230893) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0009874 (0.00211314) | 0.0000000 (0.00000000) | 0.0007800 (0.00135100)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0009700 (0.00213416) | 0.0008200 (0.00115966) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 105 | 0.0180160 (0.04024029) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0042550 (0.00972955) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0023250 (0.00398039) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 15 | 0.0032181 (0.01085890) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0056398 (0.01706862) | 0.0012400 (0.00135765) | 0.0008933 (0.00154730)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0021729 (0.00454334) | 0.0000000 (0.00000000) | 0.0002303 (0.00039895)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 105 | 0.0000094 (0.00002102) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0064197 (0.01469896) | 0.0000000 (0.00000000) | 0.0002230 (0.00038625)
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0016022 (0.00296454) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 15 | 0.0015550 (0.00250835) | 0.0000000 (0.00000000) | 0.0012000 (0.00207846)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 30 (Month 1) | 0.0085133 (0.03027644) | 0.0000000 (0.00000000) | 0.0016367 (0.00283479)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 90 (Month 3) | 0.0036457 (0.01124294) | 0.0000000 (0.00000000) | 0.0009000 (0.00155885)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 105 | 0.0010662 (0.00230033) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0008033 (0.00139141)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4) | 0.0041225 (0.00963517) | 0.0000000 (0.00000000) | 0.0018367 (0.00318120)
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12) | 0.0012100 (0.00158071) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 15 | 0.0021547 (0.00463731) | 0.0000000 (0.00000000) | 0.0034367 (0.00324179)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1) | 0.0165321 (0.03349865) | 0.0011350 (0.00160513) | 0.0035200 (0.00304882)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3) | 0.0106266 (0.01670632) | 0.0000000 (0.00000000) | 0.0038233 (0.00332250)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 105 | 0.0031980 (0.00289504) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0010800 (0.00187061)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4) | 0.0050200 (0.00831467) | 0.0000000 (0.00000000) | 0.0018300 (0.00316965)
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12) | 0.0022100 (0.00348368) | 0.0030800 (NA) — SD was not estimable for a single participant. | 0.0035050 (0.00495682)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 15 | 0.0041307 (0.00810849) | 0.0025350 (0.00091217) | 0.0033267 (0.00357693)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 30 (Month 1) | 0.0233062 (0.04002720) | 0.0185000 (0.00777817) | 0.0058683 (0.00636956)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 90 (Month 3) | 0.0169390 (0.03074260) | 0.0085000 (0.01202082) | 0.0062367 (0.00856318)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 105 | 0.0045183 (0.00427166) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0046667 (0.00808290)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4) | 0.0146317 (0.02786861) | 0.0055000 (0.00777817) | 0.0018967 (0.00184717)
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12) | 0.0047727 (0.00882216) | 0.0089800 (NA) — SD was not estimable for a single participant. | 0.0006650 (0.00094045)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 15 | 0.0046910 (0.00688923) | 0.0000000 (0.00000000) | 0.0007403 (0.00074504)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 30 (Month 1) | 0.0375398 (0.08260377) | 0.0105000 (0.01484924) | 0.0037760 (0.00368127)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 90 (Month 3) | 0.0233700 (0.04004137) | 0.0054650 (0.00176070) | 0.0013300 (0.00135044)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 105 | 0.0066317 (0.00614863) | 0.0026400 (NA) — SD was not estimable for a single participant. | 0.0005333 (0.00092376)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4) | 0.0185150 (0.03662069) | 0.0045000 (0.00636396) | 0.0015990 (0.00101474)
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12) | 0.0123264 (0.02486600) | 0.0031200 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 15 | 0.0004213 (0.00110644) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1) | 0.0004506 (0.00101312) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3) | 0.0009306 (0.00314498) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 105 | 0.0032000 (0.00715542) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4) | 0.0010313 (0.00198803) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12) | 0.0003888 (0.00109955) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 15 | 0.0033314 (0.01348231) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1) | 0.0037375 (0.01220309) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3) | 0.0020895 (0.00598185) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 105 | 0.0001374 (0.00030724) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4) | 0.0027273 (0.00904534) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12) | 0.0007944 (0.00238333) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 15 | 0.0127219 (0.01763276) | 0.0130000 (0.01838478) | 0.0251227 (0.03459943)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.1050295 (0.20473645) | 0.0500000 (0.07071068) | 0.0724367 (0.10037912)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0778682 (0.14369053) | 0.0325000 (0.04596194) | 0.0842333 (0.14123712)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 105 | 0.0423867 (0.04081753) | 0.0013300 (NA) — SD was not estimable for a single participant. | 0.0353100 (0.05329149)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0899900 (0.12840170) | 0.0433650 (0.06132737) | 0.1106733 (0.17709757)
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.1513091 (0.21942879) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0108285 (0.01438467)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 15 | 0.0509037 (0.10340779) | 0.0475000 (0.06717514) | 0.2024327 (0.30965583)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.1922011 (0.32578940) | 0.0861200 (0.11862423) | 0.2125000 (0.20614012)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.1737812 (0.29061637) | 0.1272350 (0.17361593) | 0.2045333 (0.26081536)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 105 | 0.1034720 (0.10489211) | 0.0026600 (NA) — SD was not estimable for a single participant. | 0.1804967 (0.22221367)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.1805500 (0.26929623) | 0.1188100 (0.16393564) | 0.2122567 (0.28717008)
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.1934944 (0.22273972) | 0.0030800 (NA) — SD was not estimable for a single participant. | 0.2921435 (0.39194010)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 15 | 0.0559643 (0.06460712) | 0.3345000 (0.38961584) | 0.1204393 (0.09431396)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.3096533 (0.30258266) | 1.7050000 (2.10010714) | 0.4185000 (0.53648089)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.3367906 (0.39199700) | 1.3950000 (1.81726443) | 0.4077633 (0.53498698)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 105 | 0.1848933 (0.10624645) | 0.1200000 (NA) — SD was not estimable for a single participant. | 0.2482033 (0.29841232)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.4698942 (0.59554812) | 1.4208650 (1.91465424) | 0.2656767 (0.28387658)
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.3919327 (0.07020651) | 0.0840000 (NA) — SD was not estimable for a single participant. | 0.0696435 (0.07020651)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 15 | 0.0577929 (0.07400744) | 0.1345000 (0.16334167) | 0.0337727 (0.01914939)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.4733376 (0.74274218) | 0.8520000 (1.15682669) | 0.1478333 (0.11273901)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.4983025 (0.59609158) | 0.8565000 (1.19288914) | 0.1278067 (0.11606138)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 105 | 0.3420600 (0.35216040) | 0.0250000 (NA) — SD was not estimable for a single participant. | 0.0825367 (0.07078845)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.6520608 (1.02666427) | 0.9169950 (1.28373115) | 0.1260100 (0.08686409)
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.5487509 (0.61534681) | 0.0370000 (NA) — SD was not estimable for a single participant. | 0.0216435 (0.00898945)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 15 | 0.0018039 (0.00272657) | 0.0009250 (0.00130815) | 0.0011667 (0.00202073)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0043176 (0.00745474) | 0.0086150 (0.00337290) | 0.0041833 (0.00218836)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0365866 (0.13503691) | 0.0105000 (0.01484924) | 0.0013533 (0.00117309)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 105 | 0.0321340 (0.06596445) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0021467 (0.00199362)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0212825 (0.04543103) | 0.0087300 (NA) — SD was not estimable for a single participant. | 0.0020933 (0.00313690)
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0078913 (0.01390167) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0025400 (0.00359210)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 15 | 0.0084024 (0.02103704) | 0.0042950 (0.00607405) | 0.0026897 (0.00335374)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0400210 (0.12804631) | 0.0171950 (0.01810900) | 0.0093150 (0.01317661)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0304975 (0.07184977) | 0.0080000 (0.01131371) | 0.0027633 (0.00478623)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 105 | 0.0108580 (0.01167522) | 0.0027500 (NA) — SD was not estimable for a single participant. | 0.0049600 (0.00751799)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0512582 (0.13375503) | 0.0078650 (0.01112279) | 0.0045967 (0.00557157)
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0308133 (0.07834697) | 0.0030300 (NA) — SD was not estimable for a single participant. | 0.0026885 (0.00176989)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 15 | 0.0122389 (0.01635494) | 0.0070000 (0.00989949) | 0.0557333 (0.06982874)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 30 (Month 1) | 0.1276062 (0.23983604) | 0.0304150 (0.04005760) | 0.0969917 (0.10487019)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 90 (Month 3) | 0.0542124 (0.11503390) | 0.0071500 (0.01011163) | 0.0521167 (0.07641460)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 105 | 0.0434533 (0.06315100) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0259533 (0.03276050)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 120 (Month 4) | 0.0605858 (0.09889217) | 0.0070000 (0.00989949) | 0.0488133 (0.05397085)
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS1, Day 360 (Month 12) | 0.0296555 (0.03699595) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0032750 (0.00269408)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 15 | 0.0444316 (0.07748289) | 0.0130000 (0.01838478) | 0.0280367 (0.03627084)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 30 (Month 1) | 0.3801521 (0.67068473) | 0.0512350 (0.06293957) | 0.0415883 (0.03264917)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 90 (Month 3) | 0.1645845 (0.33473334) | 0.0448850 (0.05715544) | 0.0257167 (0.01956887)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 105 | 0.1067160 (0.18769742) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0320700 (0.03599368)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 120 (Month 4) | 0.1580330 (0.28256426) | 0.0249450 (0.03119048) | 0.0141700 (0.01698637)
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS2/4, Day 360 (Month 12) | 0.0614767 (0.11059188) | 0.0030800 (NA) — SD was not estimable for a single participant. | 0.0240000 (0.03394113)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 15 | 0.0470239 (0.06626524) | 0.1770000 (0.11737973) | 0.1204000 (0.08449249)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 30 (Month 1) | 0.3655695 (0.32065242) | 0.7938700 (0.68429552) | 0.1697217 (0.15709417)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 90 (Month 3) | 0.1878077 (0.16247089) | 0.3366500 (0.37002898) | 0.0923333 (0.09666609)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 105 | 0.2131617 (0.26290060) | 0.0650000 (NA) — SD was not estimable for a single participant. | 0.0487367 (0.03451214)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 120 (Month 4) | 0.2064808 (0.20421574) | 0.2475000 (0.27223611) | 0.0493700 (0.03374277)
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS3, Day 360 (Month 12) | 0.0857582 (0.08578152) | 0.0630000 (NA) — SD was not estimable for a single participant. | 0.0191600 (0.01674429)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 15 | 0.0506306 (0.07605994) | 0.0575000 (0.05727565) | 0.0524000 (0.01247678)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 30 (Month 1) | 0.4990933 (0.64014167) | 0.3928700 (0.50186197) | 0.1050550 (0.03026614)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 90 (Month 3) | 0.2820981 (0.37844969) | 0.1433750 (0.19081276) | 0.0326667 (0.01106044)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 105 | 0.1576200 (0.17541417) | 0.0092500 (NA) — SD was not estimable for a single participant. | 0.0218933 (0.02273292)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 120 (Month 4) | 0.2221475 (0.32806338) | 0.1045000 (0.12091526) | 0.0220367 (0.00571385)
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, NS5, Day 360 (Month 12) | 0.1124982 (0.16603829) | 0.0062300 (NA) — SD was not estimable for a single participant. | 0.0027100 (0.00186676)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 15 | 0.0020544 (0.00530875) | 0.0000000 (0.00000000) | 0.0033700 (0.00583701)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 30 (Month 1) | 0.0057029 (0.01291375) | 0.0010400 (0.00147078) | 0.0006167 (0.00106810)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 90 (Month 3) | 0.0476683 (0.19290073) | 0.0000000 (0.00000000) | 0.0002203 (0.00038163)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 105 | 0.0042000 (0.00939149) | 0.0011900 (NA) — SD was not estimable for a single participant. | 0.0004167 (0.00072169)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 120 (Month 4) | 0.0031775 (0.00663800) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0003180 (0.00033860)
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, C, Day 360 (Month 12) | 0.0023488 (0.00154967) | 0.0062500 (NA) — SD was not estimable for a single participant. | 0.0005100 (0.00072125)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 15 | 0.0178773 (0.06036485) | 0.0035250 (0.00229810) | 0.0024100 (0.00301442)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 30 (Month 1) | 0.0834539 (0.27160793) | 0.0172600 (0.01199253) | 0.0023883 (0.00272227)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 90 (Month 3) | 0.0340990 (0.08904184) | 0.0061500 (0.00281428) | 0.0009000 (0.00155885)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 105 | 0.0072940 (0.00965853) | 0.0055000 (NA) — SD was not estimable for a single participant. | 0.0006200 (0.00107387)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 120 (Month 4) | 0.0588364 (0.17313721) | 0.0000000 (0.00000000) | 0.0005067 (0.00072507)
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-2, prME, Day 360 (Month 12) | 0.0090167 (0.02159530) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 15 | 0.0003586 (0.00095429) | 0.0000000 (0.00000000) | 0.0003867 (0.00066973)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0012376 (0.00387489) | 0.0000400 (0.00005657) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0002343 (0.00074914) | 0.0009350 (0.00132229) | 0.0109367 (0.01894286)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 105 | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0038700 (0.00670304)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0017572 (0.00350183) | 0.0000000 (0.00000000) | 0.0040167 (0.00695707)
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0005464 (0.00126041) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 15 | 0.0008511 (0.00168955) | 0.0008500 (0.00120208) | 0.0033333 (0.00577350)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0005805 (0.00114013) | 0.0023600 (0.00333754) | 0.0004017 (0.00055503)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0004906 (0.00099670) | 0.0000000 (0.00000000) | 0.0073200 (0.01007451)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 105 | 0.0007740 (0.00154767) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0011780 (0.00287673) | 0.0000000 (0.00000000) | 0.0035633 (0.00463250)
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0023900 (0.00325169) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0102150 (0.00596091)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 15 | 0.0004690 (0.00108044) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0008031 (0.00199994) | 0.0047450 (0.00671044) | 0.0028333 (0.00490748)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0010852 (0.00176370) | 0.0022150 (0.00313248) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 105 | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0007067 (0.00122398)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0003138 (0.00073427) | 0.0000000 (0.00000000) | 0.0113500 (0.01026974)
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0009045 (0.00166618) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 15 | 0.0010010 (0.00144763) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0012721 (0.00302348) | 0.0000450 (0.00006364) | 0.0000467 (0.00008083)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0018919 (0.00612723) | 0.0016550 (0.00234052) | 0.0059367 (0.01028261)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 105 | 0.0000050 (0.00001225) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.0005142 (0.00121641) | 0.0015450 (0.00218496) | 0.0070000 (0.01212436)
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0016991 (0.00376328) | 0.0000400 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 15 | 0.0003723 (0.00107549) | 0.0000000 (0.00000000) | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0008947 (0.00141229) | 0.0065000 (0.00919239) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0001547 (0.00044269) | 0.0000000 (0.00000000) | 0.0061467 (0.00600538)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 105 | 0.0108000 (0.01819890) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0037833 (0.01041435) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0083333 (0.01443376)
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0074013 (0.01825981) | 0.0000400 (NA) — SD was not estimable for a single participant. | 0.0277150 (0.01515330)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 15 | 0.0004090 (0.00081029) | 0.0000000 (0.00000000) | 0.0170000 (0.02944486)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0004844 (0.00107834) | 0.0000000 (0.00000000) | 0.0002883 (0.00049941)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0003021 (0.00109132) | 0.0007600 (0.00107480) | 0.0118367 (0.01821354)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 105 | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0004136 (0.00137188) | 0.0000000 (0.00000000) | 0.0053333 (0.00923760)
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0011589 (0.00257448) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0377150 (0.01030255)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 15 | 0.0028214 (0.00421069) | 0.0020000 (0.00282843) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 30 (Month 1) | 0.0046852 (0.00622110) | 0.0000000 (0.00000000) | 0.0040000 (0.00458258)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 90 (Month 3) | 0.0014295 (0.00279758) | 0.0040000 (0.00565685) | 0.0023333 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 105 | 0.0010000 (0.00200000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0070000 (0.00888819)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 120 (Month 4) | 0.0030000 (0.00441073) | 0.0010000 (0.00141421) | 0.0003333 (0.00057735)
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS1, Day 360 (Month 12) | 0.0044918 (0.00731866) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0060000 (0.00848528)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 15 | 0.0058100 (0.00997299) | 0.0025000 (0.00353553) | 0.0053333 (0.00378594)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 30 (Month 1) | 0.0049679 (0.00700541) | 0.0015000 (0.00212132) | 0.0020000 (0.00346410)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 90 (Month 3) | 0.0030861 (0.00437015) | 0.0010000 (0.00141421) | 0.0046667 (0.00808290)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 105 | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0053333 (0.00757188)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 120 (Month 4) | 0.0040000 (0.00418994) | 0.0000000 (0.00000000) | 0.0093333 (0.01137248)
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS2/4, Day 360 (Month 12) | 0.0084900 (0.00839871) | 0.0060000 (NA) — SD was not estimable for a single participant. | 0.0120000 (0.00707107)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 15 | 0.0031157 (0.00523026) | 0.0010000 (0.00141421) | 0.0010000 (0.00173205)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 30 (Month 1) | 0.0031300 (0.00536305) | 0.0000000 (0.00000000) | 0.0070000 (0.00500000)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 90 (Month 3) | 0.0029057 (0.00488854) | 0.0075000 (0.01060660) | 0.0013333 (0.00230940)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 105 | 0.0010000 (0.00244949) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0013333 (0.00230940)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 120 (Month 4) | 0.0011667 (0.00251661) | 0.0000000 (0.00000000) | 0.0036667 (0.00635085)
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS3, Day 360 (Month 12) | 0.0050373 (0.00755522) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0080000 (0.00000000)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 15 | 0.0020662 (0.00415237) | 0.0025000 (0.00353553) | 0.0050000 (0.00458258)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 30 (Month 1) | 0.0043576 (0.00713583) | 0.0000000 (0.00000000) | 0.0060000 (0.00600000)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 90 (Month 3) | 0.0020010 (0.00385930) | 0.0035000 (0.00494975) | 0.0023333 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 105 | 0.0016667 (0.00265832) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0053333 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 120 (Month 4) | 0.0040000 (0.00529150) | 0.0040000 (0.00565685) | 0.0066667 (0.01154701)
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, NS5, Day 360 (Month 12) | 0.0015591 (0.00239132) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0070000 (0.00848528)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 15 | 0.0152389 (0.04708044) | 0.0090000 (0.01272792) | 0.0033333 (0.00577350)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 30 (Month 1) | 0.0052506 (0.00585230) | 0.0000000 (0.00000000) | 0.0023333 (0.00208167)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 90 (Month 3) | 0.0044441 (0.00551617) | 0.0195000 (0.01060660) | 0.0043333 (0.00750555)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 105 | 0.0078000 (0.01744133) | 0.0090000 (NA) — SD was not estimable for a single participant. | 0.0013333 (0.00115470)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 120 (Month 4) | 0.0076250 (0.01245492) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0023333 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, C, Day 360 (Month 12) | 0.0159263 (0.01687248) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0095000 (0.01060660)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 15 | 0.0039386 (0.00920362) | 0.0000000 (0.00000000) | 0.0043333 (0.00585947)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 30 (Month 1) | 0.0042890 (0.00519741) | 0.0000000 (0.00000000) | 0.0040000 (0.00692820)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 90 (Month 3) | 0.0037368 (0.00647081) | 0.0000000 (0.00000000) | 0.0033333 (0.00577350)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 105 | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0056667 (0.00737111)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 120 (Month 4) | 0.0032727 (0.00392660) | 0.0020000 (0.00282843) | 0.0013333 (0.00230940)
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-2, prME, Day 360 (Month 12) | 0.0063789 (0.00762607) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0045000 (0.00494975)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 15 | 0.0058029 (0.01553300) | 0.0060000 (0.00848528) | 0.0126667 (0.02193931)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 30 (Month 1) | 0.0103476 (0.01374186) | 0.0090000 (0.00848528) | 0.0400000 (0.06928203)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 90 (Month 3) | 0.0141552 (0.02722292) | 0.0070000 (0.00989949) | 0.0426667 (0.06379133)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 105 | 0.0141667 (0.02123598) | 0.0270000 (NA) — SD was not estimable for a single participant. | 0.0533333 (0.06880649)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 120 (Month 4) | 0.0327508 (0.05413463) | 0.0385000 (0.01484924) | 0.0526667 (0.09122134)
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS1, Day 360 (Month 12) | 0.0594618 (0.09358403) | 0.0030000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 15: number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 15 | 0.0188947 (0.02597596) | 0.1070000 (0.13293607) | 0.2126667 (0.24855851)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 30 (Month 1) | 0.0218395 (0.03032141) | 0.0555000 (0.06010408) | 0.2116667 (0.21159946)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3): number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 90 (Month 3) | 0.0217506 (0.03474512) | 0.0770000 (0.10889444) | 0.2006667 (0.22830097)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 105 | 0.0232000 (0.01003494) | 0.0150000 (NA) — SD was not estimable for a single participant. | 0.1756667 (0.14911181)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4): number analyzed (Participants) | 10 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 120 (Month 4) | 0.0698280 (0.11664297) | 0.1095000 (0.13930004) | 0.1763333 (0.25602799)
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS2/4, Day 360 (Month 12) | 0.0789200 (0.08581529) | 0.0180000 (NA) — SD was not estimable for a single participant. | 0.2550000 (0.34648232)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 15 | 0.0101905 (0.01632825) | 0.0415000 (0.02616295) | 0.0160000 (0.01969772)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 30 (Month 1) | 0.0269048 (0.03805993) | 0.3430000 (0.33234019) | 0.1503333 (0.19894807)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 90 (Month 3) | 0.0510614 (0.06214111) | 0.3680000 (0.5176021) | 0.1486667 (0.20771455)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 105 | 0.0508333 (0.05468242) | 0.1040000 (NA) — SD was not estimable for a single participant. | 0.1286667 (0.16850618)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 120 (Month 4) | 0.0494400 (0.05523830) | 0.5175000 (0.67952962) | 0.1460000 (0.21915291)
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS3, Day 360 (Month 12) | 0.0526782 (0.05324075) | 0.0530000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 15 | 0.0088638 (0.01482118) | 0.0350000 (0.02262742) | 0.0426667 (0.05021288)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 30 (Month 1) | 0.0344576 (0.03851547) | 0.0780000 (0.05656854) | 0.0683333 (0.08251263)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 90 (Month 3) | 0.0603471 (0.11313845) | 0.0870000 (0.12303658) | 0.0323333 (0.01778576)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 105: number analyzed (Participants) | 6 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 105 | 0.0643333 (0.09686004) | 0.0410000 (NA) — SD was not estimable for a single participant. | 0.0390000 (0.00871780)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4): number analyzed (Participants) | 12 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 120 (Month 4) | 0.0471067 (0.06000386) | 0.0940000 (0.11879394) | 0.0090000 (0.01558846)
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12): number analyzed (Participants) | 11 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, NS5, Day 360 (Month 12) | 0.0758600 (0.11250364) | 0.0090000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 15: number analyzed (Participants) | 18 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 15 | 0.0103350 (0.01602034) | 0.0230000 (0.00000000) | 0.0760000 (0.06919538)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 30 (Month 1) | 0.0085812 (0.01180887) | 0.0285000 (0.00777817) | 0.0773333 (0.06971609)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3): number analyzed (Participants) | 17 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 90 (Month 3) | 0.0198388 (0.04371084) | 0.0065000 (0.00919239) | 0.0423333 (0.03516153)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 105 | 0.0380000 (0.05251190) | 0.0100000 (NA) — SD was not estimable for a single participant. | 0.0653333 (0.06033517)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4): number analyzed (Participants) | 8 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 120 (Month 4) | 0.0123363 (0.01514560) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0233333 (0.01527525)
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12): number analyzed (Participants) | 8 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, C, Day 360 (Month 12) | 0.0363138 (0.05384733) | 0.0440000 (NA) — SD was not estimable for a single participant. | 0.0050000 (0.00707107)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 15 | 0.0054286 (0.00981311) | 0.0110000 (0.00141421) | 0.0326667 (0.04051337)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 30 (Month 1) | 0.0054275 (0.00814845) | 0.0130000 (0.00141421) | 0.0266667 (0.04618802)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 90 (Month 3) | 0.0091942 (0.01593313) | 0.0165000 (0.02333452) | 0.0060000 (0.01039230)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 105 | 0.0174000 (0.01399286) | 0.0080000 (NA) — SD was not estimable for a single participant. | 0.0080000 (0.01216553)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 120 (Month 4) | 0.0141164 (0.02282460) | 0.0350000 (0.03818377) | 0.0000000 (0.00000000)
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-2, prME, Day 360 (Month 12) | 0.0237878 (0.03150909) | 0.0080000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 15 | 0.0066860 (0.01511548) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0120563 (0.02306468) | 0.0000650 (0.00009192) | 0.0008400 (0.00145492)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0025821 (0.00448167) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 105 | 0.0009780 (0.00177382) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0007567 (0.00131059)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0114040 (0.01887834) | 0.0008900 (0.00125865) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0016822 (0.00344548) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 15 | 0.0030476 (0.01094264) | 0.0000000 (0.00000000) | 0.0011667 (0.00202073)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1) | 0.0076840 (0.01657770) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3) | 0.0023789 (0.00539609) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 105 | 0.0012082 (0.00231967) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4) | 0.0042031 (0.01075305) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12) | 0.0001489 (0.00044667) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 15 | 0.0184242 (0.02939174) | 0.0089250 (0.00717713) | 0.0051230 (0.00771231)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0591005 (0.11403676) | 0.0210900 (0.02391435) | 0.0164220 (0.01587121)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0313922 (0.04328981) | 0.0190000 (0.02687006) | 0.0114300 (0.01150064)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 105 | 0.0078900 (0.00938985) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0081933 (0.00716934)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0976318 (0.16524353) | 0.0153650 (0.02172939) | 0.0053067 (0.00378127)
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0295267 (0.04211372) | 0.0029900 (NA) — SD was not estimable for a single participant. | 0.0051685 (0.00321239)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 15 | 0.0220818 (0.05553037) | 0.0025100 (0.00083439) | 0.0020167 (0.00122676)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 30 (Month 1) | 0.1106415 (0.28502664) | 0.0203700 (0.01466539) | 0.0049517 (0.00371622)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 90 (Month 3) | 0.0434985 (0.10671828) | 0.0063250 (0.00279307) | 0.0043667 (0.00583981)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 105 | 0.0047020 (0.00507315) | 0.0052300 (NA) — SD was not estimable for a single participant. | 0.0020467 (0.00354493)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 120 (Month 4) | 0.0668900 (0.14991991) | 0.0060000 (0.00848528) | 0.0072167 (0.00913589)
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-3, prME, Day 360 (Month 12) | 0.0047733 (0.00369270) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0007200 (0.00101823)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 15 | 0.0001975 (0.00067344) | 0.0015500 (0.00219203) | 0.0064300 (0.00844954)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0006700 (0.00147478) | 0.0011950 (0.00168999) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0004426 (0.00153225) | 0.0000000 (0.00000000) | 0.0106033 (0.01836551)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 105 | 0.0001760 (0.00039355) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0006105 (0.00166994) | 0.0014550 (0.00205768) | 0.0050000 (0.00556776)
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0016056 (0.00247607) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0097150 (0.01373908)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 15 | 0.0031952 (0.00507926) | 0.0000000 (0.00000000) | 0.0056667 (0.00550757)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 30 (Month 1) | 0.0049365 (0.00709962) | 0.0000000 (0.00000000) | 0.0036667 (0.00404145)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 90 (Month 3) | 0.0043447 (0.00780649) | 0.0040000 (0.00000000) | 0.0046667 (0.00568624)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 105 | 0.0052000 (0.00589067) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0050000 (0.00624500)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 120 (Month 4) | 0.0027273 (0.00405194) | 0.0065000 (0.00919239) | 0.0073333 (0.00945163)
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-3, prME, Day 360 (Month 12) | 0.0067122 (0.00782834) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0045000 (0.00212132)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 15 | 0.0090000 (0.01403916) | 0.0255000 (0.00494975) | 0.0260000 (0.04503332)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 30 (Month 1) | 0.0099805 (0.01591483) | 0.0205000 (0.01343503) | 0.0383333 (0.04645787)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 90 (Month 3) | 0.0107505 (0.01922024) | 0.0205000 (0.02899138) | 0.0056667 (0.00513160)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 105 | 0.0202000 (0.02198181) | 0.0070000 (NA) — SD was not estimable for a single participant. | 0.0130000 (0.01473092)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 120 (Month 4) | 0.0142545 (0.01922025) | 0.0440000 (0.06222540) | 0.0120000 (0.02078461)
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-3, prME, Day 360 (Month 12) | 0.0427178 (0.07626460) | 0.0050000 (NA) — SD was not estimable for a single participant. | 0.0150000 (0.02121320)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 15 | 0.0014671 (0.00263630) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0026483 (0.00397803) | 0.0020800 (0.00294156) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0018358 (0.00385801) | 0.0016100 (0.00227688) | 0.0002253 (0.00039029)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 105 | 0.0000000 (0.00000000) | 0.0027000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0008555 (0.00283722) | 0.0008400 (0.00118794) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0039322 (0.00916710) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 15 | 0.0003738 (0.00092592) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1) | 0.0009323 (0.00205020) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3) | 0.0003679 (0.00110265) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 105 | 0.0000000 (0.00000000) | 0.0027000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4) | 0.0002582 (0.00058436) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12) | 0.0002267 (0.00068000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 15 | 0.0103743 (0.01256981) | 0.0017750 (0.00019092) | 0.0052593 (0.00613561)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0138195 (0.01653836) | 0.0125800 (0.01190768) | 0.0101350 (0.00905302)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0082212 (0.01488787) | 0.0048250 (0.00682358) | 0.0045720 (0.00505935)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 105 | 0.0066820 (0.00839444) | 0.0150000 (NA) — SD was not estimable for a single participant. | 0.0066967 (0.00634139)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0150073 (0.01487729) | 0.0162450 (0.01058539) | 0.0029540 (0.00453868)
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0149633 (0.02271217) | 0.0058400 (NA) — SD was not estimable for a single participant. | 0.0170000 (0.02404163)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 15 | 0.0059200 (0.01028071) | 0.0036850 (0.00289207) | 0.0002477 (0.00042897)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 30 (Month 1) | 0.0154140 (0.02895635) | 0.0261500 (0.02807214) | 0.0023900 (0.00272666)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 90 (Month 3) | 0.0076211 (0.01271810) | 0.0046900 (0.00005657) | 0.0020187 (0.00116433)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 105 | 0.0061340 (0.00559455) | 0.0081100 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 120 (Month 4) | 0.0059764 (0.00713827) | 0.0037600 (0.00294156) | 0.0009700 (0.00149362)
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg+, IL2-, TNFa-, DENV-4, prME, Day 360 (Month 12) | 0.0034878 (0.00469261) | 0.0029200 (NA) — SD was not estimable for a single participant. | 0.0004985 (0.00070499)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 15 | 0.0006238 (0.00118351) | 0.0016350 (0.00231224) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0003618 (0.00078989) | 0.0000350 (0.00004950) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0005989 (0.00122750) | 0.0000000 (0.00000000) | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 105 | 0.0000000 (0.00000000) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0000000 (0.00000000)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0012515 (0.00280308) | 0.0014600 (0.00206475) | 0.0053333 (0.00923760)
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0005133 (0.00152134) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0047150 (0.00666802)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 15 | 0.0048171 (0.00860057) | 0.0060000 (0.00848528) | 0.0046667 (0.00416333)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 30 (Month 1) | 0.0068115 (0.00782670) | 0.0000000 (0.00000000) | 0.0026667 (0.00461880)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 90 (Month 3) | 0.0027321 (0.00433336) | 0.0050000 (0.00707107) | 0.0006667 (0.00115470)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 105 | 0.0000000 (0.00000000) | 0.0080000 (NA) — SD was not estimable for a single participant. | 0.0076667 (0.00929157)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 120 (Month 4) | 0.0023636 (0.00273030) | 0.0060000 (0.00848528) | 0.0123333 (0.01721434)
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2+, TNFa-, DENV-4, prME, Day 360 (Month 12) | 0.0080456 (0.00651373) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0050000 (0.00565685)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 15 | 0.0157619 (0.02615375) | 0.0595000 (0.05868986) | 0.1193333 (0.06900242)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1): number analyzed (Participants) | 20 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 30 (Month 1) | 0.0130950 (0.01958094) | 0.0180000 (0.02545584) | 0.0733333 (0.09451631)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3): number analyzed (Participants) | 19 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 90 (Month 3) | 0.0124347 (0.01836407) | 0.0125000 (0.01767767) | 0.0330000 (0.02868798)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 105: number analyzed (Participants) | 5 | 1 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 105 | 0.0238000 (0.02763512) | 0.0240000 (NA) — SD was not estimable for a single participant. | 0.0176667 (0.01703917)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4): number analyzed (Participants) | 11 | 2 | 3
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 120 (Month 4) | 0.0106618 (0.01504292) | 0.0300000 (0.03535534) | 0.0293333 (0.05080682)
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12): number analyzed (Participants) | 9 | 1 | 2
  IFNg-, IL2-, TNFa+, DENV-4, prME, Day 360 (Month 12) | 0.0337200 (0.04946269) | 0.0000000 (NA) — SD was not estimable for a single participant. | 0.0800000 (0.11313708)

15. Secondary Outcome: Percentage of Participants With Vaccine Viremia for Each of the Four Vaccine Strains After Vaccination
Description: Vaccine viremia was assessed for each of the four vaccine strain serotypes: TDV-1, TDV-2, TDV-3 and TDV-4. Vaccine viral ribonucleic acid (RNA) was detected by a quantitative reverse transcription-polymerase chain reaction (qRT-PCR) assay. Percentages were rounded off to the nearest decimal place.
Time Frame: Days 6, 9, 12, 15, 30 (Month 1), 90 (Month 3), 96, 99, 102, 105, 120 (Month 4)
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccine. One participant was seropositive for all dengue strains at Screening and was therefore not allocated to dengue serotype 1 or 3 positive groups. The participant did receive two vaccine doses and was thus included in Safety Analysis Set. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Unassigned Group: One participant did not meet the randomization criteria and was not allocated to any of the arm groups and was excluded from all analyses except safety analysis.
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 1
percentage of participants
  Day 6: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 6: TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 33.3 [0.8 to 90.6] | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 6: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 6: TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 9: TDV-1: number analyzed (Participants) | 21 | 4 | 3 | 1
  Day 9: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 9: TDV-2: number analyzed (Participants) | 21 | 4 | 3 | 1
  Day 9: TDV-2 | 19.0 [5.4 to 41.9] | 75.0 [19.4 to 99.4] | 66.7 [9.4 to 99.2] | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 9: TDV-3: number analyzed (Participants) | 21 | 4 | 3 | 1
  Day 9: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 9: TDV-4: number analyzed (Participants) | 21 | 4 | 3 | 1
  Day 9: TDV-4 | 4.8 [0.1 to 23.8] | 25.0 [0.6 to 80.6] | 33.3 [0.8 to 90.6] | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 12: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 12: TDV-2: number analyzed (Participants) | 22 | 4 | 2 | 1
  Day 12: TDV-2 | 50.0 [28.2 to 71.8] | 25.0 [0.6 to 80.6] | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 12: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 12: TDV-4 | 4.5 [0.1 to 22.8] | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 15: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 15: TDV-2 | 36.4 [17.2 to 59.3] | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 15: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 15: TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 30 (Month 1): TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 30 (Month 1): TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 30 (Month 1): TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 30 (Month 1): TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 90 (Month 3): TDV-1: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 90 (Month 3): TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 90 (Month 3): TDV-2: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 90 (Month 3): TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 90 (Month 3): TDV-3: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 90 (Month 3): TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 90 (Month 3): TDV-4: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 90 (Month 3): TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 96: TDV-1: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 96: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 96: TDV-2: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 96: TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 96: TDV-3: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 96: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 96: TDV-4: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 96: TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 99: TDV-1: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 99: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 99: TDV-2: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 99: TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 99: TDV-3: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 99: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 99: TDV-4: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 99: TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 102: TDV-1: number analyzed (Participants) | 21 | 3 | 3 | 1
  Day 102: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 102: TDV-2: number analyzed (Participants) | 21 | 3 | 3 | 1
  Day 102: TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 102: TDV-3: number analyzed (Participants) | 21 | 3 | 3 | 1
  Day 102: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 102: TDV-4: number analyzed (Participants) | 21 | 3 | 3 | 1
  Day 102: TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 105: TDV-1: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 105: TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 105: TDV-2: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 105: TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 105: TDV-3: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 105: TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 105: TDV-4: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 105: TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 120 (Month 4): TDV-1: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 120 (Month 4): TDV-1 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 120 (Month 4): TDV-2: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 120 (Month 4): TDV-2 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 120 (Month 4): TDV-3: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 120 (Month 4): TDV-3 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.
  Day 120 (Month 4): TDV-4: number analyzed (Participants) | 22 | 3 | 3 | 1
  Day 120 (Month 4): TDV-4 | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia. | 0.0 [NA to NA] — The 95% CI was not estimable as no participants had vaccine viremia.

16. Secondary Outcome: Duration of Vaccine Viremia for Each of the Four Vaccine Strains After Vaccination
Description: The duration of vaccine viremia for each vaccine strain was defined as the date when vaccine viremia was last detected (positive result) to date when vaccine viremia was first detected (positive result) + 1 day. It was assessed for each of the four vaccine strains: TDV-1, TDV-2, TDV-3 and TDV-4. Vaccine viral RNA was detected by qRT-PCR assay. Safety Analysis Set included all participants who received at least 1 dose of trial vaccine.
Time Frame: Up to Day 120 (Month 4)
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccine. One participant was seropositive for all dengue strains at Screening and was therefore not allocated to dengue serotype 1 or 3 positive groups. The participant did receive two vaccine doses and was thus included in Safety Analysis Set. Overall number analyzed=participants with data available for analyses. Number analyzed= participants with data available for analysis for the specified category.
Measure: Median (Full Range); unit: days
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 14 | 4 | 3 | 0
days
  TDV-2: number analyzed (Participants) | 13 | 3 | 2 | 0
  TDV-2 | 4.0 [1 to 8] | 1.0 [1 to 2] | 2.5 [1 to 4] |
  TDV-4: number analyzed (Participants) | 1 | 1 | 1 | 0
  TDV-4 | 3.0 [3 to 3] | 1.0 [1 to 1] | 1.0 [1 to 1] |

17. Secondary Outcome: Level of Vaccine Viremia for Each of the Four Vaccine Strains After Vaccination
Description: Vaccine viremia was assessed for each of the four vaccine strain serotypes: TDV-1, TDV-2, TDV-3 and TDV-4. Vaccine viral RNA was detected by qRT-PCR assay.
Time Frame: Days 6, 9, 12, and 15
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: log10 of genome equivalent per mL
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 0
log10 of genome equivalent per mL
  Day 6: TDV-1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 6: TDV-2: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 6: TDV-2 |  |  | 3.17 (NA) — SD was not estimable for a single participant. |
  Day 6: TDV-3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 6: TDV-4: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 9: TDV-1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 9: TDV-2: number analyzed (Participants) | 4 | 3 | 2 | 0
  Day 9: TDV-2 | 3.46 (0.485) | 3.94 (0.568) | 4.06 (1.003) |
  Day 9: TDV-3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 9: TDV-4: number analyzed (Participants) | 1 | 1 | 1 | 0
  Day 9: TDV-4 | 3.98 (NA) — SD was not estimable for a single participant. | 3.90 (NA) — SD was not estimable for a single participant. | 3.71 (NA) — SD was not estimable for a single participant. |
  Day 12: TDV-1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 12: TDV-2: number analyzed (Participants) | 11 | 1 | 0 | 0
  Day 12: TDV-2 | 3.43 (0.140) | 3.65 (NA) — SD was not estimable for a single participant. |  |
  Day 12: TDV-3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 12: TDV-4: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 12: TDV-4 | 3.80 (NA) — SD was not estimable for a single participant. |  |  |
  Day 15: TDV-1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 15: TDV-2: number analyzed (Participants) | 8 | 0 | 0 | 0
  Day 15: TDV-2 | 3.32 (0.172) |  |  |
  Day 15: TDV-3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Day 15: TDV-4: number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Reactions Following Each Vaccination
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included injection site pain [Grade 0 (no pain), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity with or without treatment) and 3 (severe: prevents daily activity with or without treatment)], injection site erythema [Grade 0 (<25 mm), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)] and injection site swelling [Grade 0 (<25 mm), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)]. Only categories for which there was at least 1 participant are reported.
Time Frame: Within 7 days after each of the vaccine dose given on Day 1 (Month 0) and 90 (Month 3)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 1
percentage of participants
  After First Vaccination: Any Solicited Local AEs | 54.5 | 25.0 | 66.7 | 0
  After First Vaccination: Pain | 40.9 | 25.0 | 66.7 | 0
  After First Vaccination: Erythema | 40.9 | 0 | 33.3 | 0
  After Second Vaccination: Any Solicited Local AEs: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Any Solicited Local AEs | 68.2 | 50.0 | 66.7 | 0
  After Second Vaccination: Pain: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Pain | 59.1 | 50.0 | 66.7 | 0
  After Second Vaccination: Erythema: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Erythema | 31.8 | 0 | 33.3 | 0
  After Second Vaccination: Swelling: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Swelling | 9.1 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Solicited Systemic Reactions Following Each Vaccination
Description: Solicited systemic AEs were collected by participants using diary cards within 14 days after vaccination and will include fever, headache, asthenia, malaise and myalgia. Severity grades are: Grade 0: none, Grade 1: mild (no interference with daily activity), Grade 2: moderate (interference with daily activity with or without treatment), Grade 3: severe (prevents normal daily activity with or without treatment). A systemic AE of fever (defined as body temperature ≥ 100.4°F regardless of method taken) was derived from a daily temperature reading recorded within 14 days after vaccination. Only categories for which there was at least 1 participant are reported.
Time Frame: Within 14 days after each of the vaccine dose given on Day 1 (Month 0) and 90 (Month 3)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 1
percentage of participants
  After First Vaccination: Any Solicited Systemic AE | 68.2 | 75.0 | 100.0 | 0
  After First Vaccination: Headache | 50.0 | 50.0 | 33.3 | 0
  After First Vaccination: Myalgia | 40.9 | 25.0 | 100.0 | 0
  After First Vaccination: Asthenia | 31.8 | 25.0 | 66.7 | 0
  After First Vaccination: Malaise | 54.5 | 25.0 | 100.0 | 0
  After First Vaccination: Fever | 4.5 | 0 | 0 | 0
  After Second Vaccination: Any Solicited Systemic AE: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Any Solicited Systemic AE | 27.3 | 0 | 66.7 | 0
  After Second Vaccination: Headache: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Headache | 13.6 | 0 | 66.7 | 0
  After Second Vaccination: Myalgia: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Myalgia | 9.1 | 0 | 0 | 0
  After Second Vaccination: Asthenia: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Asthenia | 18.2 | 0 | 0 | 0
  After Second Vaccination: Malaise: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination: Malaise | 13.6 | 0 | 66.7 | 0

20. Secondary Outcome: Percentage of Participants With at Least One Unsolicited Adverse Events (AEs) Following Each Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a study vaccine; it does not necessarily have to have a causal relationship with study vaccine administration.
Time Frame: Up to 28 days (day of vaccination + 27 days) after administration of each vaccine dose given on Day 1 (Month 0) and 90 (Month 3)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 1
percentage of participants
  After First Vaccination | 63.6 | 75.0 | 66.7 | 0
  After Second Vaccination: number analyzed (Participants) | 22 | 2 | 3 | 1
  After Second Vaccination | 36.4 | 0 | 100.0 | 0

21. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A SAE is defined as any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or / significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the aforementioned criteria.
Time Frame: From first vaccination (Day 1) through end of study (Day 360 [Month 12])
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccine. One participant was seropositive for all dengue strains at Screening and was therefore not allocated to dengue serotype 1 or 3 positive groups. The participant did receive two vaccine doses and was thus included in Safety Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 1
percentage of participants | 4.5 | 25.0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With Medically Attended AEs (MAAEs)
Description: MAAEs was defined as AEs leading to a medical visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From first vaccination (Day 1) through end of study (Day 360 [Month 12])
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
Number analyzed (Participants) | 22 | 4 | 3 | 1
percentage of participants | 45.5 | 50.0 | 33.3 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious Adverse Events: From first vaccination through end of study (Day 360 [Month 12]); Non-serious (Other) AEs: Up to 28 days (day of vaccination + 27 days) after administration of each vaccine dose on Day 1 [Month 0] and Day 90 [Month 3]
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Safety Analysis Set included all participants who received at least one dose of trial vaccine. One participant was seropositive for all dengue strains at Screening and was therefore not allocated to dengue serotype 1 or 3 positive groups. The participant did receive two vaccine doses and was thus included in Safety Analysis Set.
Arm/Group | TDV: Flavivirus-naïve | TDV: DENV Immune: DENV-1 Positive | TDV: DENV Immune: DENV-3 Positive | Unassigned Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/4 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/4 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 22/22 | 4/4 | 3/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDV: Flavivirus-naïve (N=22) | TDV: DENV Immune: DENV-1 Positive (N=4) | TDV: DENV Immune: DENV-3 Positive (N=3) | Unassigned Group (N=1)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDV: Flavivirus-naïve (N=22) | TDV: DENV Immune: DENV-1 Positive (N=4) | TDV: DENV Immune: DENV-3 Positive (N=3) | Unassigned Group (N=1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 9 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 13 | 1 | 2 | 0
Eye pain (Eye disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 14 | 2 | 2 | 0
Injection site bruising (General disorders) | 1 | 1 | 1 | 0
Injection site pruritus (General disorders) | 2 | 0 | 0 | 0
Malaise (General disorders) | 13 | 1 | 3 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pain (General disorders) | 15 | 1 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Swelling (General disorders) | 8 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 5 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03746015/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT03746015/SAP_002.pdf